

# Protocol No. MC2-01-C3 Novella Study No. NYA14539

#### STATISTICAL ANALYSIS PLAN

A Randomised, Multicentre, Open-label, Parallel-group Maximal Use Trial, Evaluating the Pharmacokinetic Profile of the Active Ingredients and their Metabolites after Application of MC2-01 Cream Compared with Active Comparator in Subjects with Extensive Psoriasis Vulgaris

Novella Clinical 365 West Passaic Street Rochelle Park, NJ 07662, USA

21 September 2018

Version No. Amendment 1.0

Johan Selmer, MD VP Medical Affairs MC2 Therapeutics

Carol Udell, MS Sr. Director, Clinical Reporting Novella Clinical Johan Schmir

7 - Septer Name: Uoffah Seming 7 EDT
Signing Reason: Jeg godkender dette dokument
Signing Time: 21-09-2018 11:43:31 EDT

OCB84AC3A754477D9A7870027DF16AE6

Carol Udull

11-Septen 2018 ne | Carol: Udot 46 EDT

DocuSigned by:

Signing Reason: I approve this document Signing Time: 9/21/2018 12:15:36 PM EDT

-CE741CD0FE9741ECA29CB39E84B183BB

# **Table of Contents**

| 1. | INTRODUC | CTION | 5 |
|-----------|---------------|--------------------------------------|----|
| 2. | STUDY OB | BJECTIVES | 5 |
| 3. | STUDY DE | SIGN | 5 |
| 4. | | RE AND SOFTWARE | |
| <b>5.</b> | DATABASI | E CLOSURE | 7 |
| 6. | SAMPLE S | IZE DETERMINATION | 7 |
| 7. | HANDLING | G OF MISSING DATA | 7 |
| 8. | ANALYSIS | POPULATIONS | 7 |
| 9. | DATA CON | NVENTIONS FOR ANALYSIS | 8 |
| | 9.1 General | Statistical Principles | 8 |
| | 9.2 Study D | ay and Baseline | 8 |
| 10. | STATISTIC | CAL EVALUATION | 8 |
| | 10.1 Subje | ct Disposition | 8 |
| | 10.2 Proto | col Deviation | 8 |
| | 10.3 Demo | graphic and Baseline Characteristics | 9 |
| | 10.4 Study | Drug Exposure and Accountability | 9 |
| | 10.5 Prior | and Concomitant Medications | 10 |
| | 10.6 Concu | urrent Procedures | 10 |
| | 10.7 Medic | cal History | 10 |
| | 10.8 Safety | y Analysis | 10 |
| | 10.8.1 Safety | y Endpoints | 10 |
| | 10.8.2 Analy | vses of Safety Endpoints | 11 |
| | 10.8.2.1 | HPA-axis Suppression | 11 |
| | 10.8.2.2 | Calcium Metabolism Endpoints | 12 |
| | 10.8.2.3 | Adverse Events | 12 |
| | 10.8.2.5 | Safety Laboratory Parameters | 13 |
| | 10.8.2.6 | Vital Signs | 14 |
| | 10.8.2.7 | Electrocardiograms (ECG) | 14 |
| | 10.8.3 Physic | cal Examination (PE) | 14 |
| | 10.9 Pharm | nacokinetics Analysis | 14 |
| | 10.9.1 Analy | sis of Pharmacokinetic Parameters | 14 |

| | 10.10 Ana | alysis of Other Endpoints | 16 |
|---|---|---|---|
| | 10.10.1 | Physician Global Assessment of Psoriasis Severity (PGA) | 16 |
| | 10.10.2 | Body Surface Area Involvement of Psoriasis (BSA) | 16 |
| | 10.10.3 | Psoriasis Treatment Convenience Scale (PTCS) | 16 |
| 11. | CHANGE | ES FROM THE PROTOCOL AND PLANNED ANALYSES | 16 |
| <b>12.</b> | HEADIN | GS | 18 |
| 13. | ARCHIV | ING AND RETENTION OF DOCUMENTS | 18 |
| 14. | OUTLIN | E OF PROPOSED TABLES, FIGURES AND LISTINGS | 19 |

# **List of Abbreviations and Definitions of Terms**

| Abbreviation | Definition |
|---|---|
| ACTH | Adrenocorticotropic hormone |
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| AUC <sub>0-7</sub> | Area under the time-concentration curve from time zero to 7 hours |
| AUC <sub>0-t</sub> | Area under the time-concentration curve from time zero to the last measurable concentration |
| $\mathrm{AUC}_{\scriptscriptstyle{0\text{-}\infty}}$ | Area under the time-concentration curve from time zero to infinity |
| BDP | Betamethasone dipropionate |
| BSA | Body surface area |
| CAL | Calcipotriene (United States term) / Calcipotriol (European Union term) |
| C <sub>max</sub> | Maximum plasma drug concentration |
| CRO | Contract Research Organisation |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| FDA | Food and Drug Administration |
| HPA | Hypothalamic-pituitary-adrenal |
| ICF | Informed consent form |
| IP | Investigational product |
| IRB | Institutional Review Board |
| IWR | Interactive web response |
| MCV | Mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| OTC | Over the counter |
| PGA | Physician's Global Assessment |
| PK | Pharmacokinetics |
| PTH | Parathyroid hormone |
| RBC | Red blood cell |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SOP | Standard operating procedure |
| T <sub>1/2</sub> | Elimination half-life |
| T <sub>max</sub> | Time to maximum plasma drug concentration |
| UPT | Urine pregnancy test |
| US | United States |
| WBC | White blood cell |

# 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the study Protocol version 3.0 dated December 20, 2017.

This document provides additional details concerning the statistical analyses outlined in the protocol and reflects any changes to the protocol from any amendments. This plan will not repeat all the definitions given in the protocol but will provide further details of the summaries and analyses planned therein.

#### 2. STUDY OBJECTIVES

The primary objective is to evaluate the pharmacokinetic profile of the active ingredients and their main metabolites after application of MC2-01 cream, and compare with the active comparator following once daily topical application under maximum-use conditions in subjects with extensive psoriasis vulgaris.

The secondary objective is to evaluate the effect of MC2-01 cream on the hypothalamic-pituitary-adrenal (HPA) axis and calcium metabolism following once daily topical application under maximum-use conditions in subjects with extensive psoriasis vulgaris.

# 3. STUDY DESIGN

This is a Phase 2, randomised, open-label, parallel-group, multicentre trial in which the investigational product, MC2-01 cream, and CAL/BDP ointment (comparator) are investigated in subjects with clinically diagnosed extensive psoriasis vulgaris of disease severity assessed by Physician's Global Assessment (PGA) of at least moderate (Figure 1). Subjects who meet inclusion/exclusion criteria will be randomly assigned in a 1:1 ratio to receive either MC2-01 cream or the comparator. Subjects assigned to MC2-01 cream will apply 1 dose of trial medication topically once daily for 8 weeks and the subjects assigned to the comparator will apply 1 dose of trial medication topically once daily for 4 weeks.

At Week 4, the pharmacokinetic (PK) profile of calcipotriene (CAL), betamethasone dipropionate (BDP) and their main metabolites MC1080 and betamethasone 17-propionate, respectively, will be assessed for both treatment groups. At Week 8, the PK profile of CAL, BDP and their main metabolites will be assessed for the MC2-01 cream treatment group only. At Week 4 and Week 8, the effect of once-daily use of MC2-01 cream on the HPA axis and calcium metabolism will be evaluated for MC2-01 cream treatment group. Other safety assessments (local skin reactions, AEs, laboratory tests, electrocardiogram (ECG)), vital signs and physical examinations) and efficacy assessments are also performed.

Figure 1: Study Design

#### Trial Design for Subjects Assigned to the MC2-01 Cream



<sup>\*</sup>Follow-up visits will be required only for subjects who have unresolved AEs or whose calcium levels have not returned to pretreatment levels at the End of Treatment visit.

#### Trial Design for Subjects Assigned to the Active Comparator



<sup>\*</sup>Follow-up visits will be required only for subjects who have unresolved AEs at the End of Treatment visit.

#### 4. HARDWARE AND SOFTWARE

Statistical analysis will be performed following Novella Clinical standard operating procedures (SOP) and on the Novella Clinical computer network. All statistical analysis will be performed using SAS Version 9.3 or higher with program code prepared specifically for the project by qualified Novella Clinical statisticians and SAS programmers.

The SAS programs will generate rich-text-formatted (RTF) output with the "RTF" extension using the SAS Output Delivery System (ODS). The summary tables and listings will be formatted using the Times New Roman 9-point font. The RTF output is included in report documents prepared with Microsoft Word and converted to PDF format without typographical change.

Study data tabulation model (SDTM) data sets and analysis data model (ADaM) data sets will be created and taken as input to validated SAS programs to generate the report-ready tables, listings,

and figures. Each output display will show the names of the data sets and SAS program used to produce it.

#### 5. DATABASE CLOSURE

After completion of all data review procedures, validation of the project database, and approval of the data review document by the study sponsor, the clinical database will be closed. Any change to the clinical database after this time will require written authorization, with explanation, by the Sponsor and the Biostatistician.

#### 6. SAMPLE SIZE DETERMINATION

The choice of sample size in this trial is not based on statistical considerations, but rather on regulatory considerations with respect to common practice in maximum use studies evaluating pharmacokinetic profiles and evidence of HPA safety. The chosen number of approximately 25 subjects included in the PK population at Week 4 in each treatment arm is considered sufficient to compare the PK properties corresponding to the two treatments.

#### 7. HANDLING OF MISSING DATA

No imputation will be made for missing data.

# 8. ANALYSIS POPULATIONS

Three analysis populations will be defined for analysis:

- <u>Safety Population</u>: will include all randomized subjects who have been dispensed the trial medication, excluding subjects who return all of the trial medication unopened. The Safety Population will be used for all safety analyses other than evaluation of the HPAaxis.
- HPA population: will include all subjects in the Safety population that are assigned to MC2-01 cream and who show normal HPA function at Baseline (defined as a 30-minute post-stimulation cortisol level ≥18 μg/dL). Since the objective of the analysis is to estimate the risk to subjects with normal HPA function of HPA-axis suppression following treatment, subjects who meet the definition of HPA-axis suppression at Baseline will be excluded from the analysis. The HPA population will be used for the HPA axis suppression analysis.
- <u>Pharmacokinetic (PK) Population:</u> will include all subjects in the Safety population who have received the planned application of treatment at the Week 4 or Week 8 visit, respectively, and have had at least one post-application blood draw for PK assessment at the corresponding visit. The PK Population will be used for the PK analysis.

All safety, HPA and PK analyses will be conducted according to the treatment actually received.

#### 9. DATA CONVENTIONS FOR ANALYSIS

#### 9.1 General Statistical Principles

All statistical processing will be performed using the SAS system (Version 9.3 or higher).

All observed and derived variables (e.g., change from baseline) used in the summaries of analyses will be presented in by-subject listings. Descriptive statistics will be used to provide an overview of the safety and PK results. For categorical parameters, the number and percentage of subjects in each category will be presented. The denominator for percentage will be based on the number of subjects appropriate for the purpose of analysis. For continuous parameters, descriptive statistics will include number of observations, mean, standard deviation (SD), median, and range. The PK parameters will be summarised using appropriate descriptive statistics including median, lower and upper quartiles, minimum and maximum. Geometric means and coefficient of variation (CV) will be provided as appropriate.

It is planned that the data from all centers that participate in this protocol will be combined so that an adequate number of subjects will be available for analysis.

No interim analyses are planned.

# 9.2 Study Day and Baseline

For purpose of the SAP, Day 1 is defined as the date of first application of study drug, which corresponds to Randomization/Visit 1 of the study protocol. Study day is calculated relative to the date of Day 1.

Baseline is defined as the last available measurement prior to first application of study drug. Change from baseline is defined as the post-baseline value minus the baseline value.

#### 10. STATISTICAL EVALUATION

#### 10.1 Subject Disposition

The number and percentage of subjects who are screened, randomized, included in each analysis population, who complete the study, and withdraw from the study (overall and by reason for withdrawal) will be summarized, overall and by treatment group.

A by-subject enrolment and disposition listing will be presented for all randomized subjects.

#### 10.2 Protocol Deviation

Protocol deviations will be presented in a by-subject listing.

#### 10.3 Demographic and Baseline Characteristics

Demographics, baseline characteristics will be summarized overall and by treatment for the Safety, HPA and PK populations. The following demographic and baseline variables will be included:

- Age (years)
- Gender
- Race
- Ethnicity
- Fitzpatrick Skin Type
- Weight (kg)
- Height (cm)
- Baseline HPA Axis Suppression Status (MC2-01 cream group only)
- Baseline PGA
- Baseline Total BSA (%)
- Duration of psoriasis in years (calculated as year of baseline minus year of first psoriasis diagnosis)

#### 10.4 Study Drug Exposure and Accountability

Subjects will record the date of each trial medication application in the subject diary. The kit number, and corresponding date dispensed and returned will be collected.

The weight of the returned kits will also be collected.

The following parameters of study medication exposure will be summarized by treatment group and by study period, i.e., from day 1 to Week 4 (both groups) and from day 1 to Week 8 (MC2-01 cream group), for the Safety Population:

- Total number of days of exposure to the study drug, defined as the date of last application of study drug during the period minus date of first application plus one. The last application is the in-clinic dosing at Week 4 visit (Day 1 to Week 4 period) and Week 8 visit (Day 1 to Week 8 period).
- Total number of missed doses during each study period per subject diary
- Total number of applications during each study period, defined as the total number of doses
  required minus total number of doses missed. Total number of required doses is defined as
  total number of days of exposure minus any days of investigator approved stop (if
  applicable)
- Total weight of trial medication used (g) during each study period, defined as the summation of amount of drug used for all dispensed kits. Amount of drug used per kit is defined as the difference in weight between the returned and dispensed kits, where weight

of dispensed kits is a unit value. Amount of drug used for sealed and unreturned kits will be assumed to be  $0.0~\mathrm{g}$ 

• Amount of drug used per week (g/per week), defined as the total amount of drug used divided by total number of days of exposure to the study drug multiplied by 7

#### 10.5 Prior and Concomitant Medications

Prior (with stop dates prior to Day 1) and concomitant medications (ongoing or with stop dates on or after Day 1) for all randomised subjects will be provided in a by-subject listing. Concomitant medications will be summarized by WHO-DDE Anatomical-Therapeutic-Chemical (ATC) classification and preferred term (PT) for each treatment for Safety population.

For the determination of prior vs. concomitant medications, the following rules regarding the stop date will be applied:

- If only year was recorded, and it is before Day 1, it is a prior medication; if year is same or after Day 1, it is assumed to be a concomitant medication.
- If day is missing, but month and year are before Day 1, it is a prior medication; if month and year are the same or after Day 1, it is assumed to be a concomitant medication.
- If start date is after Day 1, it is a concomitant medication regardless.

Psoriasis treatment history will be displayed in a by-subject listing.

#### **10.6** Concurrent Procedures

All concurrent procedures will be provided in a by subject listing for all randomized subjects.

#### **10.7** Medical History

Past and current medical conditions will be coded using MedDRA dictionary (version 20.0). Medical history for all randomized subjects will be provided in a by-subject listing.

#### 10.8 Safety Analysis

#### **10.8.1 Safety Endpoints**

Primary safety endpoints include:

• HPA-axis suppression

HPA-axis function will be assessed in a challenge test with an intravenous dose of adrenocorticotropic hormone (ACTH) (Cosyntropin). **Normal HPA function** is, based on the Cosyntropin US Packing Insert (USPI) (revision May 2018), defined as a 30-minute post-stimulation cortisol level  $\geq$ 18 µg/dL.

Conversely, **HPA-axis suppression** is defined as 30-minute post-stimulation cortisol level <18 µg/dL.

HPA-axis function status will be considered as missing if post-stimulation serum cortisol level is missing.

- Changes in calcium metabolism endpoints from 24-hour urinalysis, including
  - o Albumin-corrected serum calcium
  - o 24 hours urinary calcium excretion
  - o Ratio of urinary calcium to creatinine

# Other safety endpoints include:

- Adverse events (AEs)
- Local Skin Reaction (LSR) Assessment
  - o Investigator assessed signs: erythema, scaling, edema, atrophy, vesicles and erosion/ulceration; vesicles, and erosion/ulceration
  - O Subject assessed symptoms: burning or pain
- Laboratory parameters
  - Hematology: hemoglobin, hematocrit, red blood cell (RBC) count, mean corpuscular volume (MCV), white blood cell (WBC) count, including differential count and platelet count.
  - Serum biochemistry: cortisol, urea, glucose, creatinine, calcium, albumin, calcium (albumin corrected), sodium, potassium, chloride, calcium, phosphate, alkaline phosphatase (ALP), plasma parathyroid hormone (PTH), 25-OH Vitamin D (Visit 1 only)
  - o 24-hour urinalysis: calcium, phosphate, creatinine, volume, total calcium excretion, total phosphate excretion, total creatinine excretion, urinary calcium:creatinine ratio, urinary phosphate:creatinine ratio
- Vital signs (blood pressure, pulse rate)
- Standard 12-lead electrocardiogram (ECG) (MC2-01 cream subjects only)
- Physical examination (PE)

# 10.8.2 Analyses of Safety Endpoints

#### 10.8.2.1 HPA-axis Suppression

The number and proportion of subjects with HPA-axis suppression at Week 4 will be summarised for the HPA population. Subjects with HPA-axis suppression at Week 4, was as described in the

protocol, contacted to discontinue use of MC2-01 cream. Subjects with HPA-axis suppression at Week 8 will be summarised overall and separately by HPA-axis suppression status at Week 4.

An additional analysis of the number and proportion of subjects with HPA-axis suppression will be summarised based on the test laboratory normal reference range established for the analytical method used by the test laboratory in the trial for the ACTH challenge test.

• In this analysis HPA suppression is defined as a 30-minute post-stimulation cortisol level < 14  $\mu g/dl$  (test laboratory normal reference range of 14 to 36  $\mu g/dl$  for the 30-minute post-stimulation cortisol level). This analysis will be performed among MC2-01 cream subjects whose Baseline cortisol level is  $\geq$  14  $\mu g/dl$ 

All HPA-axis function test results (baseline, Week 4, Week 8, and Follow-up) will be presented in a by-subject listing for the Safety population.

#### 10.8.2.2 Calcium Metabolism Endpoints

All calcium metabolism data will be presented in a by-subject listing for the following parameters:

- Albumin-corrected serum calcium
- 24 hours urinary calcium excretion
- Ratio of urinary calcium to creatinine

Observed values and changes from baseline to Week 4 and Week 8 will be summarized using descriptive statistics for subjects in the Safety population assigned to MC2-01 cream.

#### 10.8.2.3 Adverse Events

AE terms will be coded using MedDRA dictionary (version 20.0). A treatment-emergent AE (TEAE) is defined as an AE with a start date on or after the first application to trial medication (Day 1). If relationship to study medication is missing, the event will be conservatively summarized as being related to study drug. If intensity is missing, a separate category of missing intensity will be included in the summary table, and no imputation of severity will be performed. Through the data cleaning process, all attempts will be made to avoid missing values for relationship and severity.

All AEs will be presented in a by-subject listing, detailing the verbatim term given by the investigator, the PT, SOC, whether or not related to Cosyntropin or study procedure, location of AE to treatment area, start date, stop date, intensity, outcome, relationship to study medication (definitely, probably, possibly, and not related), action taken with study medication, action taken to treat the AE, seriousness and criteria for seriousness. For subjects assigned to MC2-01 cream, all TEAEs will be assigned to the Week 1-4 (starting from Day 1 to 28) or post-Week 4 period (starting from Day 29 and after) based on onset dates. Serious AEs and AEs leading to study drug discontinuation will be presented in a separate listing.

An overall summary of AEs will be presented by treatment and by period (MC2-01 group only). The summary will include the total number of events, frequency counts and percentages with:

- Any AE
- Any TEAE
- Any serious TEAE
- Any treatment-related TEAE
- Any TEAE leading to study drug discontinuation

Summaries of the incidence of TEAEs will be displayed by treatment and by period (MC2-01 group only) according to the following:

- All TEAEs by PT in descending order of frequency (the combined frequency of both treatments)
- All TEAEs by SOC, PT, and maximum severity (mild, moderate, or severe)
- All TEAEs by SOC, PT, and maximum relationship (recorded as 'definitely', 'probably', and 'possibly') to the study drug

At each level of summarization, a subject will be counted once if he/she reported one or more events. The severity of TEAEs and relationship to study drug will be summarized in a similar manner. For summaries of relationship to study drug, a subject will be classified according to the closest relationship. For summaries of TEAE severity, a subject will be classified according to the highest severity.

# 10.8.2.4 Local Skin Reaction (LSR) Assessment

LSR assessments by investigator and subject will be summarized using frequency counts and percentages by treatment and visit. By-subject listings will be provided.

#### **10.8.2.5** Safety Laboratory Parameters

Clinical laboratory (hematology, biochemistry and urinalysis) results will be presented in bysubject listings. Abnormal laboratory findings will be flagged and presented in a separate listing.

Absolute values, changes from baseline, and relative changes from baseline (defined as ratio of the post-baseline vs baseline value) will be summarized using descriptive statistics (means, medians, standard deviations, ranges, and coefficient of variations) by treatment and by visit. Shift tables using extended normal ranges (baseline to Week 4 and most extreme post-baseline value up to Week 4 for both arms) will also be provided.

Urine pregnancy test will be presented in a by-subject listing for subjects with childbearing potential.

#### **10.8.2.6** Vital Signs

Vital signs data will be presented in a by-subject listing. Observed values and changes from baseline will be summarized using descriptive statistics by treatment and visit.

#### 10.8.2.7 Electrocardiograms (ECG)

ECG data will be presented in a by-subject listing, with flagging of abnormal results.

# 10.8.3 Physical Examination (PE)

Physical examination results will be present in a by-subject listing.

#### 10.9 Pharmacokinetics Analysis

All analyses of pharmacokinetics (PK) will be based on the PK population.

All available concentration results will be summarised using appropriate descriptive statistics (number of subjects, number of quantifiable concentrations, median, lower and upper quartiles, minimum, maximum) for active ingredients (BDP and CAL) and for their major metabolites. A listing for sample date/times as well as derived sampling time deviations will be provided. Median and individual concentration versus time curves will be plotted (linear and semi-log plots). Nominal sample collection times will be used in determining concentration descriptive statistics and plotting median concentration versus time profiles.

All analyte concentrations below the lower limit of quantification (BLOQ) will be reported as the lower limit of quantification (LLoQ) and will be treated as LLoQ in descriptive statistics and plasma concentration-time profiles.

#### 10.9.1 Analysis of Pharmacokinetic Parameters

Plasma PK parameters shown below (AUC<sub>0-t</sub>, AUC<sub>0- $\infty$ </sub>, AUC<sub>0- $\infty$ </sub>, AUC<sub>0-7</sub>, C<sub>max</sub>, T<sub>max</sub>, and T<sub>½</sub>) will be calculated at Week 4 in subjects randomized to comparator and MC2-01 groups and Week 8 in subjects randomized to MC2-01 cream only.

For a given analyte, the PK parameters  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ ,  $T_{max}$ , and  $T_{\frac{1}{2}}$  will be calculated if data allow.  $AUC_{0-7}$  and  $C_{max}$  will be calculated using standard formulas inserting the lower limit of quantification (LLoQ) for non-quantifiable levels of the analyte; therefore,  $AUC_{0-7}$  will be an upper limit in case at least one time point shows a non-quantifiable level of the analyte, and  $C_{max}$  will be an upper limit in case all time points show non-quantifiable levels of the analyte.

| $C_{max}$ | Maximum plasma drug concentration. BLOQ Concentrations will be |
|-----------|----------------------------------------------------------------|
| | treated as LLoQ for this calculation |

| T <sub>max</sub> | Time to maximum plasma drug concentration. If the maximum concentration value occurs at more than one time point, $T_{\text{max}}$ is defined as the first time point with this value |
|---|---|
| AUC <sub>0-7</sub> | Area under the time-concentration curve from time zero to 7 hours, as calculated by the linear trapezoidal method. BLOQ Concentrations will be treated as LLoQ for this calculation |
| AUC <sub>0-t</sub> | Area under the time-concentration curve from time zero to the last quantifiable concentration |
| AUC <sub>0-∞</sub> | Area under the time-concentration curve from time zero to infinity, calculated as $AUC_{0-t} + C_{tf}/\lambda z$ , where $C_{tf}$ is the last concentration $\geq LoQ$ . $AUC_{0-\infty}$ will be calculated only if $\lambda z$ can be calculated. |
| T <sub>1/2</sub> | Elimination half-life, calculated as $ln(2)/\lambda z$ . $T_{1/2}$ will not be calculated if $\lambda z$ cannot be determined |
| Λz | Elimination (terminal phase) rate constant, calculated as the slope of the terminal phase linear regression line of the log-scale concentration over the time points corresponding to the elimination phase of the concentration-time profiles. The elimination rate constant, $\lambda z$ , will not be calculated if the elimination phase of the log-linear concentration-time profile cannot be fit with an appropriate regression line. The time points corresponding to a subject's elimination phase will be identified by visually examining the log-scale concentration-time profile. A minimum of three points, not including $C_{max}$ , in which there is a relatively straight downward trend in concentration when plotted on a log scale, and the adjusted $R^2$ value for the fitted line must be at least 0.9 is required for the determination of $\lambda z$ . As an additional confirmation of the suitability of $\lambda z$ , the log-linear profile, which includes the regression line through the terminal points, will be checked via visual inspection, to determine whether the regression appropriately represents the terminal slope. |

PK parameters will be listed and summarized using descriptive statistics (n, median, lower and upper quartiles, minimum and maximum) where appropriate. Geometric means and geometric CV will be calculated for  $AUC_{0-1}$ ,  $AUC_{0-\infty}$ ,  $AUC_{0-7}$ , and  $C_{max}$  as appropriate. An exception to this is  $T_{max}$  and  $T_{\frac{1}{2}}$  where only median, minimum, and maximum will be presented.

Assessment of systemic exposure (Week 4)

Novella No. NYA14539

Assessment of relative systemic exposure in the two treatment arms will be performed for AUC<sub>0-7</sub> and C<sub>max</sub> at Week 4. If any of the post-dose time point shows a non quantifiable level of the analyte, the calculated PK parameters will be considered left censored. In particular, AUC<sub>0-7</sub> will be considered censored if at least one post-dose concentration is below LLOQ. C<sub>max</sub> will be considered censored if all post-dose values are below LLOQ. To account for the censored data, the SAS PROC LIFEREG procedure will be used on log-transformed PK parameters with treatment group as a fixed effect. Geometric mean ratio and associated 90% confidence interval (CI) (back-transformed from the estimates) will be presented.

# 10.10 Analysis of Other Endpoints

#### 10.10.1Physician Global Assessment of Psoriasis Severity (PGA)

PGA will be summarised using frequency counts and percentages for each treatment at Week 4 (all subjects) and at Week 8 (subjects assigned to MC2-01 cream). The proportion of subjects with treatment success, defined as a minimum 2-point decrease from Baseline in the PGA will also be summarized.

#### 10.10.2Body Surface Area Involvement of Psoriasis (BSA)

BSA results will be presented in a by-subject listing.

#### 10.10.3 Psoriasis Treatment Convenience Scale (PTCS)

The PTCS consists of 6 disease-specific, self-report questions with a recall period of 1 week and rated on a 1-10 scale.

- 1. How easy was the treatment to apply to the skin?
- 2. How greasy was the treatment when applying it to the skin?
- 3. How moisturised did your skin feel after applying the treatment?
- 4. How greasy did your skin feel <u>after</u> applying the treatment?
- 5. How much did treating your skin disrupt your daily routine?
- 6. Overall, how satisfied were you with the medical treatment?

Each of the questions and the sum of the first 5 questions of PTCS will be summarized using descriptive statistics by treatment for Week 4. Sum of the first 5 question will be further compared between MC2-01 cream and the active comparator using a mixed effect model with treatment as a systematic effect and study site as a random effect. Treatment difference (MC2-01 cream minus active comparator) along with 95% CI will be reported.

#### 11. CHANGES FROM THE PROTOCOL AND PLANNED ANALYSES

The 30 minutes ACTH test using the ACTH analogue tetracosactide to stimulate cortisol secretion from the adrenals is an effective test for the assessment of the HPA axis in subjects with pituitary

disease. Diagnostic criteria for adrenal insufficiency have traditionally relied both on the absolute level of cortisol 30 minutes after injection of tetracosactide as well as a requirement of an absolute increase in cortisol during the test. The diagnostic criteria used in the MC2-01-C3 protocol was based on the USPI dated February 2012 (1) for Cosyntropin in which there were specific requirements to plasma cortisol both concerning the level of increase as well as the 30 minutes value according to the original description of the test (2) when testing morning samples. The diagnostic value of an absolute increase in cortisol has, however, been challenged. Several studies, e.g.(3, 4) have shown that calculation of the increment cortisol increase is of no diagnostic value, and careful reviews (5, 6) have strongly warned against this parameter as a diagnostic criterion. As a consequence, both expert guidelines from the Endocrine Society (7) as well as the recently updated (May 2018) USPI for Cosyntropin (8) recommends the 30 minutes cortisol value as the sole diagnostic criterion for the diagnosis of adrenal insufficiency with a limit for adrenal supression of plasma cortisol < 18 μg/dl (500 nmol). This criterion is used in the evaluation of the data obtained in MC2-01-C3 trial. Furthermore, the plasma cortisol from the ACTH challenge test is measure by mass spectrometry. Mass spectrometry assays of cortisols are without any of the positive bias that plaque most cortisol immunoassays (9) and consequently limit for adrenal supression of plasma cortisol is below 14 µg/dl (390 nmol/l) according to laboratory report from the manufacturer (Quest Diagnostics) of this test. For this reason, this lower limit for plasma cortisol of 14 µg/dl (390 nmol/l) will also be used in the evaluation of the data obtained in MC2-01-C3 trial.

- 1. FDA. Cosyntropin USPI Sandoz. 2012.
- 2. Wood JB, Frankland AW, James VH, Landon J. A rapid test of adrenocortical function. Lancet. 1965;1(7379):243-5.
- 3. Patel SR, Selby C, Jeffcoate WJ. The short Synacthen test in acute hospital admissions. Clin Endocrinol (Oxf). 1991;35(3):259-61.
- 4. Widmer IE, Puder JJ, Konig C, Pargger H, Zerkowski HR, Girard J, et al. Cortisol response in relation to the severity of stress and illness. J Clin Endocrinol Metab. 2005;90(8):4579-86.
- 5. Clark PM, Neylon I, Raggatt PR, Sheppard MC, Stewart PM. Defining the normal cortisol response to the short Synacthen test: implications for the investigation of hypothalamic-pituitary disorders. Clin Endocrinol (Oxf). 1998;49(3):287-92.
- 6. Arafah BM. Hypothalamic pituitary adrenal function during critical illness: limitations of current assessment methods. J Clin Endocrinol Metab. 2006;91(10):3725-45.
- 7. Bornstein SR, Allolio B, Arlt W, Barthel A, Don-Wauchope A, Hammer GD, et al. Diagnosis and Treatment of Primary Adrenal Insufficiency: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016;101(2):364-89.

- 8. FDA. Cosyntropin USPI Sandoz. May 2018.
- 9. El-Farhan N, Pickett A, Ducroq D, Bailey C, Mitchem K, Morgan N, et al. Method-specific serum cortisol responses to the adrenocorticotrophin test: comparison of and five automated immunoassays. Clin Endocrinol (Oxf). 2013;78(5):673-80.

# 12. HEADINGS

Each page of the analysis will show the sponsor's name, the investigational product, and the protocol number. Report tables will be embedded in the MS Word report document from SAS program output without change. The footer of each table will show the name of the SAS program module which generated it, the names of all data sets providing input data in the program and the date and time the table was generated.

# 13. ARCHIVING AND RETENTION OF DOCUMENTS

After finalization of the analysis, the following will be archived at Novella Clinical and/or with the study sponsor:

- SAP and any amendments
- All SAS code used in the project for statistical analysis, report tables generation, and analysis data set creation
- Tables, listings and figures as included in the clinical study report
- SAS study data tabulation model (SDTM) and analysis dataset model (ADaM) datasets

# 14. OUTLINE OF PROPOSED TABLES, FIGURES AND LISTINGS

#### **Summary Tables**

| 14.1 | Summary of Disposition, Demographic, and Exposure Tables |
|---|---|
| 14.1.1.1 | Summary of Subject Disposition |
| 14.1.2.1 | Summary of Subject Demographics and Baseline Characteristics; Safety Population |
| 14.1.2.2 | Summary of Subject Demographics and Baseline Characteristics; HPA Population |
| 14.1.2.3 | Summary of Subject Demographics and Baseline Characteristics; PK Population |
| 14.1.3 | Summary of Extent of Exposure and Compliance; Safety Population |
| 14.1.4 | Summary of Concomitant Medications by Anatomical Therapeutic Chemical Class (ATC) and Preferred Term; Safety Population |
| 14.2 | Summary of Study Endpoints Tables |
| 14.2.1.1 | Summary of Plasma Concentration of CAL (ng/mL) by Time Point; PK Population |
| 14.2.1.2 | Summary of Plasma Concentration of BDP (ng/mL) by Time Point; PK Population |
| 14.2.1.3 | Summary of Plasma Concentration of MC1080 (ng/mL) by Time Point; PK Population |
| 14.2.1.4 | Summary of Plasma Concentration of Betamethasone 17-propionate (ng/mL) by Time Point; PK Population |
| 14.2.2.1 | Summary of Plasma Concentration of CAL (ng/mL) Pharmacokinetics Parameters; PK Population |
| 14.2.2.2 | Summary of Plasma Concentration of BDP (ng/mL) Pharmacokinetics Parameters; PK Population |
| 14.2.2.3 | Summary of Plasma Concentration of MC1080 (ng/mL) Pharmacokinetics Parameters; PK Population |
| 14.2.2.4 | Summary of Plasma Concentration of Betamethasone 17-propionate (ng/mL) Pharmacokinetics Parameters; PK Population |
| 14.2.3.1 | Assessment of Relative Systemic Exposure of CAL(ng/mL) at Week 4; PK Population |
| 14.2.3.2 | Assessment of Relative Systemic Exposure of BDP (ng/mL) at Week 4; PK Population |
| 14.2.3.3 | Assessment of Relative Systemic Exposure of MC1080 (ng/mL) at Week 4; PK Population |
| 14.2.3.4 | Assessment of Relative Systemic Exposure of Betamethasone 17-propionate (ng/mL) at Week 4; PK Population |
| 14.2.4.1 | Summary of HPA-Axis Suppression (Based on Cosyntropin US Packing Insert); HPA Population |
| 14.2.4.2 | Summary of HPA-Axis Suppression (Based on Lab Reference Range); MC2-01 Cream Subjects with Baseline Cortisol Level ≥ 14 µg/dl |
| 14.2.5 | Summary of Calcium Metabolism; HPA Population |
| 14.2.6 | Summary of Physician's Global Assessment (PGA); Safety Population |
| 14.2.7 | Summary of Psoriasis Treatment Convenience Score (PTCS) at Week 4; Safety Population |
| 14.3 | Summary of Safety Tables |
| 14.3.1.1 | Overall Summary of Adverse Events; Safety Population |
| 14.3.1.2 | Summary of Treatment-emergent Adverse Events, Weeks 1-4 by System Organ Class and Preferred Term in Descending Frequency; Safety Population |
| 14.3.1.3 | Summary of Treatment-emergent Adverse Events, Weeks 1-4 by System Organ Class, Preferred Term, and Maximum Severity; Safety Population |
| 14.3.1.4 | Summary of Treatment-emergent Adverse Events, Weeks 1-4 by System Organ Class, Preferred Term, and Maximum Causality; Safety Population |
| 14.3.2.1.1 | Summary of Clinical Laboratory Results by Treatment and Visit, Biochemistry; Safety Population |
| 14.3.2.1.2 | Summary of Clinical Laboratory Results by Treatment and Visit, Hematology; Safety Population |
| 14.3.2.2.1 | Clinical Laboratory Results, Shifts from Baseline, Biochemistry; Safety Population |
| 14.3.2.2.2 | Clinical Laboratory Results, Shifts from Baseline, Hematology; Safety Population |
| 14.3.3 | Summary of Vital Signs by Treatment and Visit; Safety Population |
| 14.3.4 | Summary of Investigator Assessed Local Skin Reactions (LSR); Safety Population |

| 14.3.5 | Summary of Subject Assessed Local Skin Reactions (LSR); Safety Population |
|---|---|
|---|---|

# **Figures**

| 14.4.1.1.1.1 | CAL Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling |
|---|---|
| 14.4.1.1.1.2 | CAL Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling CAL Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling |
| 14.4.1.1.2.1 | BDP Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling |
| 14.4.1.1.2.2 | BDP Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling |
| 14.4.1.1.3.1 | MC1080Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling |
| 14.4.1.1.3.2 | MC1080Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling MC1080Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling |
| 14.4.1.1.4.1 | Betamethasone 17-propionate Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling |
| 14.4.1.1.4.2 | Betamethasone 17-propionate Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling |
| 14.4.1.2.1.1 | CAL Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling |
| 14.4.1.2.1.2 | CAL Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling CAL Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |
| 14.4.1.2.2.1 | BDP Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |
| 14.4.1.2.2.2 | BDP Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling BDP Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |
| 14.4.1.2.3.1 | MC1080Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling |
| 14.4.1.2.3.2 | MC1080Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |
| 14.4.1.2.4.1 | Betamethasone 17-propionate Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling |
| 14.4.1.2.4.2 | Betamethasone 17-propionate Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |
| 14.4.2.1.1.1 | Individual CAL Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling |
| 14.4.2.1.1.2 | Individual CAL Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling |
| 14.4.2.1.2.1 | Individual BDP Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling |
| 14.4.2.1.2.2 | Individual BDP Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling |
| 14.4.2.1.3.1 | Individual MC1080Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling |
| 14.4.2.1.3.2 | Individual MC1080Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling |
| 14.4.2.1.4.1 | Individual Betamethasone 17-propionate Concentration (Median) by Time Point, Linear Scale, Week 4 Serial PK Sampling |
| 14.4.2.1.4.2 | Individual Betamethasone 17-propionate Concentration (Median) by Time Point, Linear Scale, Week 8 Serial PK Sampling |
| 14.4.2.2.1.1 | Individual CAL Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling |
| 14.4.2.2.1.2 | Individual CAL Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |
| 14.4.2.2.2.1 | Individual BDP Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling |
| 14.4.2.2.2.2 | Individual BDP Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |
| 14.4.2.2.3.1 | Individual MC1080Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling |
| 14.4.2.2.3.2 | Individual MC1080Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |
| 14.4.2.2.4.1 | Individual Betamethasone 17-propionate Concentration (Median) by Time Point, Semi-Log Scale, Week 4 Serial PK Sampling |
| 14.4.2.2.4.2 | Individual Betamethasone 17-propionate Concentration (Median) by Time Point, Semi-Log Scale, Week 8 Serial PK Sampling |

# **Listing Tables**

| 16.1.7 | Subject Enrolment and Randomization |
|----------|-------------------------------------|
| 16.2.1.1 | Screen Failure |

# MC2 Therapeutics Protocol No. MC2-01-C3 Novella No. NYA14539

| 1.5.21141.011 | |
|---|---|
| 16.2.1.2 | Subject Disposition |
| 16.2.2 | Protocol Deviations |
| 16.2.3 | Population Datasets |
| 16.2.4.1 | Demographics and Baseline Characteristics |
| 16.2.4.2 | Prior and Concomitant Medication |
| 16.2.4.3 | Concurrent Procedures |
| 16.2.4.4 | Medical or Surgical History |
| 16.2.4.5 | Psoriasis Treatment History |
| 16.2.5.1 | Study Drug Administration and Compliance |
| 16.2.5.2 | Study Drug Accountability |
| 16.2.5.3.1 | Overall Study Drug Exposure and Compliance, Day 1 to Week 4 Period |
| 16.2.5.3.2 | Overall Study Drug Exposure and Compliance, Day 1 to Week 8 Period |
| 16.2.5.4.1 | Subject Treatment Diary Card |
| 16.2.5.4.2 | Subject Food Diary |
| 16.2.6.1 | Plasma Concentration Sample Date and Time and Plasma Concentrations |
| 16.2.6.2.1 | CAL Derived Pharmacokinetics Parameters |
| 16.2.6.2.2 | BDP Derived Pharmacokinetics Parameters |
| 16.2.6.2.3 | MC1080 Derived Pharmacokinetics Parameters |
| 16.2.6.2.4 | Betamethasone 17-propionate Derived Pharmacokinetics Parameters |
| 16.2.6.3 | Physician's Global Assessment of Disease Severity (PGA) – Scalp, Trunk and/or Limbs |
| 16.2.6.4 | Investigator's Assessment of the Body Surface Area (BSA) Involvement of Psoriasis |
| 16.2.6.5 | Investigator and Subject Assessed Local Skin Reaction (LSR) |
| 16.2.6.6 | Psoriasis Treatment Convenience Scale |
| 16.2.6.7 | ACTH Challenge (<18 μg/dL.) |
| 16.2.6.7 | ACTH Challenge (<14 μg/dL.) |
| 16.2.7.1 | Adverse Events |
| 16.2.7.2 | Serious Adverse Events |
| 16.2.7.3 | Adverse Events Leading to Study Drug Discontinuation |
| 16.2.8.1 | Urine Pregnancy Test |
| 16.2.8.2.1 | Clinical Laboratory Test Results; Biochemistry |
| 16.2.8.2.2 | Clinical Laboratory Test Results; Hematology |
| 16.2.8.2.3 | Clinical Laboratory Test Results; 24 Hour Urinalysis |
| 16.2.8.3 | Laboratory Values Outside of Normal Range |
| 16.2.8.4 | Vital Signs |
| 16.2.8.5 | Physical Examinations |
| 16.2.8.6 | 12-Lead ECG Results |
| 16.2.9 | General Comments |


MC2 Therapeutics

Protocol Number: MC2-01-C3

Table 14.1.1: Summary of Subject Disposition

| | MC2-01 Cream | Active Comparator | Overall |
|---|---|---|---|
| Number of Subjects Screened | | | XX |
| Number of Subjects Randomized | XX | XX | XX |
| Number of Subjects in Safety Population, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of Subjects in HPA Population, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of Subjects in PK Population, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of Subjects Completing the Study, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of Subjects Discontinued, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Reason for Discontinuation, n (%) | | | |
| Investigator discretion | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unacceptable adverse events | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Exclusion criteria | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| HPA axis suppression at Visit 1/Day 0 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Albumin corrected serum calcium above upper limit at Visit 1/Day 0 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Trial suspended by Sponsor | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Voluntary withdrawal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other reasons | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Denominator for percentages is the number of subjects randomized.

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

Table 14.1.2.X: Summary of Subject Demographics and Baseline Characteristics [Safety Population] [HPA Population] [PK Population]

| | MC2-01 Cream | Active Comparator | Overall |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| Age (years) | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |
| Sex, n(%) | | | |
| Female | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Male | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Race, n(%) | | | |
| White | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Black or African American | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Asian | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| American Indian or Alaska Native | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Native Hawaiian or Other Pacific Islander | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other [1] | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Ethnicity, n(%) | | | |
| Hispanic or Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Hispanic or Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[1]</sup> See listing 16.2.4.1 for other races.

Table 14.1.2.X: Summary of Subject Demographics and Baseline Characteristics [Safety Population] [HPA Population] [PK Population]

| | MC2-01 Cream | Active Comparator | Overall |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| Fitzpatrick Skin Type, n(%) | | | |
| I | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| II | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| III | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <etc.></etc.> | | | |
| Height (cm) | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |
| Weight (kg) | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |

Note: Height and weight can be self-reported.

MC2 Therapeutics

Protocol Number: MC2-01-C3

Table 14.1.2.X: Summary of Subject Demographics and Baseline Characteristics [Safety Population] [HPA Population] [PK Population]

| | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline HPA Axis Suppression Status, n(%) | | | , |
| Yes | XX (XX.X) | | |
| No | XX (XX.X) | | |
| Unknown | XX (XX.X) | | |
| Baseline PGA (Scalp, Trunk and/or Limbs), n(%) | | | |
| 0 – Clear | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 – Almost clear | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 – Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 – Moderate | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| 4 – Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Baseline Total BSA (%) | XX | XX | XX |
| N | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Mean (SD) | XX.X | XX.X | XX.X |
| Median | XX, XX | XX, XX | XX, XX |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX | XX | XX |
| Duration of Psoriasis (years) [2] | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |

<sup>[2]</sup> Calculated as year of baseline minus year of first psoriasis diagnosis


MC2 Therapeutics

Protocol Number: MC2-01-C3

Calla 14.1.2. Carray of Francis of Francis of Carray Carra

Table 14.1.3: Summary of Extent of Exposure and Compliance Safety Population

| | Day 1 to Week 8 | Day 1 | to Week 4 |
|---|---|---|---|
| | MC2-01 Cream<br>(N=XX) | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) |
| Total Number of Days of Exposure[1] | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |
| Total Number of Missed Doses | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |
| Total Number of Doses Applied[2] | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |

<sup>[1]</sup> Total number of days of exposure is defined as the date of last application of study drug minus date of first application plus one. The last application is the in-clinic dosing at Week 4 visit (Day 1 to Week 4 period) and Week 8 visit (for Day 1 to Week 8 period).

<sup>[2]</sup> Total number of doses applied= total number of doses required – total number of missed doses. Total number of doses required = total number of days of exposure – any days of investigator approved stop.


MC2 Therapeutics

Protocol Number: MC2-01-C3

Table 14.1.3: Summary of Extent of Exposure and Compliance Safety Population

| | Day 1 to Week 8 | Day 1 | to Week 4 |
|---|---|---|---|
| | MC2-01 Cream<br>(N=XX) | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) |
| Cotal Amount of Drug Used (g)[3] | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X(XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |
| amount of Drug Used per Week (g/per week)[4] | | | |
| N | XX | XX | XX |
| Mean (SD) | XX.X(XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |

<sup>[3]</sup> Total amount of drug used (g) is defined as the summation of amount of drug used per kit for all returned kits. Amount of drug used per kit is the difference in weight between the returned and dispensed kits. Amount of drug used for sealed and unreturned kits will be assumed to be 0.0 g.

<sup>[4]</sup> Amount of drug used per week (g/per week) is defined as the total amount of drug used divided by total number of days of exposure to the study drug multiplied by 7.

Table 14.1.4: Summary of Concomitant Medications by Anatomical Therapeutic Chemical Class (ATC) and Preferred Term Safety Population

| | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) |
|---|---|---|
| | | , |
| Subjects with any Concomitant Medication, n (%) | XX (XX.X) | XX (XX.X) |
| << Anatomical Therapeutic Chemical Class >> | | |
| << Medication Preferred Term >> | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX |
| << Anatomical Therapeutic Chemical Class >> | | |
| << Medication Preferred Term >> | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX |
| << Medication Preferred Term >> | XXXXX | XXXXX |

Note: Any medication ongoing or with stop date on or after Day 1 is a concomitant medication. Counts reflect number of subjects in each treatment group reporting one or more prior medication that map to the WHO Drug anatomical therapeutic chemical or preferred term. A subject may be counted once only in each row of the table.

Table 14.2.1.X: Summary of Plasma Concentration of [CAL, BDP, MC1080, Betamethasone 17-propionate] (ng/mL) by Time Point PK Population

[MC2-01 Cream] [Active Compartor]

| Time Point | N | Nquant | Median | Lower, Upper Quartiles | Minimum, Maximum |
|---|---|---|---|---|---|
| Baseline | | | | | |
| Pre-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |
| Visit 2/Week 2 | | | | | |
| Pre-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |
| Visit 3/Week 4 | | | | | |
| Pre-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |
| 0.5 hours post-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |
| 1 hour post-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |
| 2 hours post-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |
| 3 hours post-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |
| 5 hours post-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |
| 7 hours post-dose | XX | XX | XX.X | XX.X, XX.X | XX.X, XX.X |

#### Visit 5/Week 8

<include all time points>

Note: Concentration below the limit of quantitation (< XX.X ng/mL) are reported as the lower limit of quantification (LLoQ) for calculating summary statistics. N<sub>quant</sub>: number of samples in the N population with quantifiable levels of analyte;

Table 14.2.2.X: Summary of [CAL, BDP, MC1080, Betamethasone 17-propionate] (ng/mL) Pharmacokinetics Parameters PK Population

| | N | Median | Lower Quartile, | Minimum, |
|------------------------------|----|--------|-----------------|--------------|
| | | | Upper Quartile | Maximum |
| Week 4 | | | | |
| MC2-01 Cream (N=XX) | | | | |
| $C_{max}$ (ng/mL) | XX | XXX.X | XXX, XXX | XXX, XXX |
| $T_{max}(h)$ | XX | XXX.X | XXX.X, XXX.X | XXX.X, XXX.X |
| $AUC_{0-7}$ (ng*h/mL) | XX | XXXX | XXX, XXX | XXX, XXX |
| $AUC_{0-t}$ (ng*h/mL) | XX | XXXX | XXX, XXX | XXX, XXX |
| $AUC_{0-\infty}(ng*h/mL)$ | XX | XXXX | XXX, XXX | XXX, XXX |
| $T_{1/2}$ (h) | XX | XXX.X | XXX.X, XXX.X | XXX.X, XXX.X |
| Active Comparator (N=XX) | | | | |
| $C_{max}$ (ng/mL) | XX | XXX.X | XXX, XXX | XXX, XXX |
| $T_{max}(h)$ | XX | XXX.X | XXX.X, XXX.X | XXX.X, XXX.X |
| $AUC_{0-7}$ (ng*h/mL) | XX | XXXX | XXX, XXX | XXX, XXX |
| $AUC_{0^{-t}}$ (ng*h/mL) | XX | XXXX | XXX, XXX | XXX, XXX |
| $AUC_{0-\infty}(ng*h/mL)$ | XX | XXXX | XXX, XXX | XXX, XXX |
| T <sub>1/2</sub> (h) | XX | XXX.X | XXX.X, XXX.X | XXX.X, XXX.X |
| Week 8 | | | | |
| MC2-01 Cream (N=XX) | | | | |
| $C_{max}$ (ng/mL) | XX | XXX.X | XXX, XXX | XXX, XXX |
| $T_{max}(h)$ | XX | XXX.X | XXX.X, XXX.X | XXX.X, XXX.X |
| $AUC_{0-7} (ng*h/mL)$ | XX | XXXX | XXX, XXX | XXX, XXX |
| AUC <sub>0-t</sub> (ng*h/mL) | XX | XXXX | XXX, XXX | XXX, XXX |
| $AUC_{0-\infty}(ng*h/mL)$ | XX | XXXX | XXX, XXX | XXX, XXX |
| T <sub>1/2</sub> (h) | XX | XXX.X | XXX.X, XXX.X | XXX.X, XXX.X |

MC2 Therapeutics

Protocol Number: MC2-01-C3

Page X of Y

Table 14.2.3.X: Assessment of Relative Systemic Exposure of [CAL, BDP, MC1080, Betamethasone 17-propionate] (ng/mL) at Week 4 PK Population

| | | Natural Log-S | Scale Difference[1] | Geometric Mea | an Ratio (GMR) [2] |
|---|---|---|---|---|---|
| | N | Estimate | 90% CI | Estimate | 90% CI |
| Cmax (ng/mL) | XX | X.XXX | X.XXX, X.XXX | X.XXX | X.XXX, X.XXX |
| AUC <sub>0</sub> -7 (ng*h/mL) | XX | X.XXX | X.XXX, X.XXX | X.XXX | X.XXX, X.XXX |

<sup>[1]</sup> Difference and the associated 90% CI (confidence interval), are estimated by using an analysis of variance model for censored data including treatment group, using log-transformed PK parameters.

<sup>[2]</sup> Geometric Mean ratio (GMR) and the associated 90% CI are back transformed point estimate and the associated 90% CI.

MC2 Therapeutics Protocol No. MC2-01-C3 Novella No. NYA14539  September 20, 2018

MC2 Therapeutics
Page X of Y
Protocol Number: MC2-01-C3

Table 14.2.4.1 Summary of HPA-Axis Suppression (Based on Cosyntropin US Packing Insert) HPA Population

| | MC2-01 Cream<br>(N=XX) |
|-----------------------------------|------------------------|
| HPA-Axis Suppression, n / N (%) | |
| Visit 3/ Week 4 | XX/XX (XX.X) |
| Visit 5/ Week 8 | XX/XX (XX.X) |
| HPA-Axis Suppressed at Week 4 | XX/XX (XX.X) |
| HPA-Axis Not Suppressed at Week 4 | XX/XX (XX.X) |

Note: HPA-axis suppression is defined as a 30-minute post-stimulation cortisol level <18 µg/dL Generated on XX/XX/XX:XXXX by XXXXX / Uses: XXXX / Reference: Data Listings XXXX

[Programming note: Denominator for Visit 5/Week 8 (Week 4 HPA-Axis Suppressed) row is subjects with HPA-Axis Suppressed at Week 8; denominator for Visit 5/Week 8 (Week 4 HPA-Axis Not Suppressed) row is subjects with HPA-Axis Suppressed at Week 8]

MC2 Therapeutics Protocol No. MC2-01-C3 Novella No. NYA14539  September 20, 2018

MC2 Therapeutics
Page X of Y
Protocol Number: MC2-01-C3

Table 14.2.4.2 Summary of HPA-Axis Suppression (Based on Lab Reference Range) MC2-01 Cream Subjects with Baseline Cortisol Level ≥ 14 μg/dl

| | MC2-01 Cream<br>(N=XX) |
|-----------------------------------|------------------------|
| HPA-Axis Suppression, n / N (%) | |
| Visit 3/ Week 4 | XX/XX (XX.X) |
| Visit 5/ Week 8 | XX/XX (XX.X) |
| HPA-Axis Suppressed at Week 4 | XX/XX (XX.X) |
| HPA-Axis Not Suppressed at Week 4 | XX/XX (XX.X) |

Note: HPA-axis suppression is defined as a 30-minute post-stimulation cortisol level <14 µg/dL Generated on XX/XX/XX:XXXX by XXXXX / Uses: XXXX / Reference: Data Listings XXXX

[Programming note: Denominator for Visit 5/Week 8 (Week 4 HPA-Axis Suppressed) row is subjects with HPA-Axis Suppressed at Week 8; denominator for Visit 5/Week 8 (Week 4 HPA-Axis Not Suppressed) row is subjects with HPA-Axis Suppressed at Week 8]

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

Table 14.2.5 Summary of Calcium Metabolism HPA Population

| | MC2-01 | MC2-01 Cream (N=XX) |
|---|---|---|
| | Observed Value | Change from Baseline |
| lbumin-Corrected Serum Calcium (unit) | | |
| Baseline | | |
| N | XX | |
| Mean (SD) | XX.X(XX.X) | |
| Median | XX.X | |
| Q1, Q3 | XX, XX | |
| Minimum, Maximum | XX, XX | |
| Visit 3/Week 4 | | |
| N | XX | XX |
| Mean (SD) | XX.X(XX.X) | XX.X (XX.X) |
| Median | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX |
| Visit 5/Week 8 | | |
| N | XX | XX |
| Mean (SD) | XX.X(XX.X) | XX.X (XX.X) |
| Median | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX |
| Minimum, Maximum | XX, XX | XX, XX |

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

Table 14.2.6: Summary of Physician's Global Assessment (PGA)
Safety Population

| | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) |
|---|---|---|
| | (IV AA) | (11 212) |
| seline | | |
| Observed Value, n (%) | | |
| N | XX | XX |
| 0 – Clear | XX (XX.X) | XX (XX.X) |
| 1 – Almost clear | XX (XX.X) | XX (XX.X) |
| 2 - Mild | XX (XX.X) | XX (XX.X) |
| 3 – Moderate | XX (XX.X) | XX (XX.X) |
| 4 – Severe | XX (XX.X) | XX(XX.X) |
| it 3/Week 4 | | |
| Observed Value, n (%) | | |
| N | XX | XX |
| 0 – Clear | XX(XX.X) | XX (XX.X) |
| <etc.></etc.> | XX (XX.X) | XX (XX.X) |
| Change From Baseline, n (%) | | |
| N | XX | XX |
| 2 = Worsen by $2$ | XX(XX.X) | XX (XX.X) |
| 1 = Worsen by $1$ | XX(XX.X) | XX (XX.X) |
| 0 = No Change | XX (XX.X) | XX (XX.X) |
| -1 = Improve by 1 | XX (XX.X) | XX (XX.X) |
| -2 = Improve by 2 | XX (XX.X) | XX (XX.X) |
| -3 = Improve by 3 | XX (XX.X) | XX (XX.X) |
| PGA Treatment Success [1] | XX (XX.X) | XX (XX.X) |

<sup>[1]</sup> PGA success is defined as a minimum 2-point decrease from Baseline in the PGA.

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

Table 14.2.6: Summary of Physician's Global Assessment (PGA)
Safety Population

| | MC2-01 Cream<br>(N=XX) | Active<br>Comparator<br>(N=XX) |
|---|---|---|
| isit 5/Week 8 | | |
| Observed Value, n (%) | | |
| N | XX | |
| 0 – Clear | XX (XX.X) | |
| <etc.></etc.> | XX (XX.X) | |
| Change From Baseline, n (%) | | |
| N | XX | |
| 2 = Worsen by $2$ | XX (XX.X) | |
| 1 = Worsen by $1$ | XX (XX.X) | |
| 0 = No Change | XX (XX.X) | |
| -1 = Improve by 1 | XX (XX.X) | |
| -2 = Improve by 2 | XX (XX.X) | |
| -3 = Improve by 3 | XX (XX.X) | |
| PGA Treatment Success [1] | XX (XX.X) | |

<sup>[1]</sup> PGA success is defined as a minimum 2-point decrease from Baseline in the PGA.
MC2 Therapeutics

Protocol Number: MC2-01-C3

Table 14.2.7: Summary of Psoriasis Treatment Convenience Score (PTCS) at Week 4
Safety Population

| | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) |
|---|---|---|
| C. 4.1 C (C | | |
| Fotal Score (Sum of Q1 to Q5) N | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X (XX.XX) | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X |
| Linear Mixed Effect Model[1] | | |
| LSM (SE) | XX.X(XX.X) | XX.X(XX.X) |
| LSM, 95% CI | XX.X, XX.X | XX.X, XX.X |
| LSM Difference (MC2-01 Cream - Active Comparator) (SE) | XX.X (XX.X) | , |
| LSM Difference, 95% CI | XX.X, XX.X | |
| 1: How easy was the treatment to apply to the skin? | | |
| N | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X |
| Continue for Q2: How greasy was the treatment when applying it to the skin? Q3: How moisturized did your skin feel after applying the treatment? Q4: How greasy did your skin feel after applying the treatment? | | |
| Q5: How much did treating your skin disrupt your daily routine? | | |
| Q6: Overall, how satisfied were you with the medical treatment?>> | | |

SE = Standard error; LSM = Least square means; CI = Confidence interval

<sup>[1]</sup> The linear mixed effect model includes as a systematic effect and study site as a random effect.

Table 14.3.1.1: Overall Summary of Adverse Events
Safety Population

| | Wee | ks 1 – 4 [1] | Post Week 4 [2] |
|---|---|---|---|
| | MC2-01 Cream<br>(N=XX) | Active Comparator<br>(N=XX) | MC2-01 Cream<br>(N=XX) |
| Adverse Events | | | |
| Number of Events | XX | XX | XX |
| Number of Subjects, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Freatment-Emergent Adverse Events (TEAEs) | | | |
| Number of Events | XX | XX | XX |
| Number of Subjects, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Γreatment-Related TEAEs | | | |
| Number of Events | XX | XX | XX |
| Number of Subjects, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Serious AEs (All) | | | |
| Number of Events | XX | XX | XX |
| Number of Subjects, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Serious TEAEs | | | |
| Number of Events | XX | XX | XX |
| Number of Subjects, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| AEs Leading to Study Drug Discontinuation | | | |
| Number of Events | XX | XX | XX |
| Number of Subjects, n (%) | XX (XX.X) | XX (XX.X) | XX(XX.X) |

Note: Counts reflect number of subjects reporting one or more adverse events that map to MedDRA 20.0. A subject will be counted once only within each AE category. TEAEs include all AEs starting or worsening after the first dose of study drug.

MC2 Therapeutics

Protocol Number: MC2-01-C3

Page X of Y

Table 14.3.1.2: Summary of Treatment-emergent Adverse Events by System Organ Class and Preferred Term in Descending Frequency Safety Population

| | Week | s 1 – 4 [1] | Post Week 4 [2] |
|---|---|---|---|
| System Organ Class<br>Preferred Term | MC2-01 Cream<br>(N=XX) | Active Comparator<br>(N=XX) | MC2-01 Cream<br>(N=XX) |
| Subjects with any TEAE, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event System Organ Class >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event System Organ Class >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA system organ class or preferred term. A subject may be counted once only in each row of the table.

<sup>[1]</sup> Includes TEAEs with an onset date on or before Week 4 visit.

<sup>[2]</sup> Includes TEAEs with an onset date after Week 4 visit.

<sup>&</sup>lt;Programming Note: sort by SOC in alphabetical order and PT in descending order of the combined frequency in the two active treatments>

MC2 Therapeutics

Protocol Number: MC2-01-C3

Table 14.3.1.3: Summary of Treatment-emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity

| by System Organ Class, Preferred Term, and Maximum Severity |
|-------------------------------------------------------------|
| Safety Population |
| Weeks 1 – 4 [ |

| | | Weel | ks 1 – 4 [1] | Post Week 4 [2] |
|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Severity | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) | MC2-01 Cream (N=XX) |
| Treicircu Term | Severity | (IV-AA) | (11-AA) | (11-AA) |
| Subjects with any TEAE, n (%) | Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event System Organ Class >> | Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Mild | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | Severe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Moderate | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Mild | XX (XX.X) | XX (XX.X) | XX(XX.X) |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA system organ class or preferred term. A subject may be counted only once at the highest severity. AEs are categorized by onset date.

MC2 Therapeutics

Protocol Number: MC2-01-C3

Table 14.3.1.4: Summary of Treatment-emergent Adverse Events by System Organ Class. Preferred Term, and Maximum Causality

by System Organ Class, Preferred Term, and Maximum Causality Safety Population

| | | Wee | Post Week 4 [2] | |
|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Causality Assessment[1] | MC2-01 Cream<br>(N=XX) | Active Comparator<br>(N=XX) | MC2-01 Cream<br>(N=XX) |
| Subjects with any TEAE, n (%) | Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Not Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event System Organ Class >> | Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Not Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| << Adverse Event Preferred Term >> | Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Not Related | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA system organ class or preferred term. A subject may be counted only once at the highest severity. AEs are categorized by onset date.

MC2 Therapeutics

Protocol Number: MC2-01-C3

Page X of Y

Table 14.3.2.1.X: Summary of Clinical Laboratory Results by Treatment and Visit

[Biochemistry][Hematology]

Safety Population

[Lab Tests Name (Units)]

| | Mo | MC2-01 Cream (N=XX) | | | Active Comparator (N=XX) | |
|---|---|---|---|---|---|---|
| | Observed Value | CFBL | Relative CFBL | Observed Value | CFBL | Relative CFBL |
| seline | | | | | | |
| N | XX | | | XX | | |
| Mean (SD) | XX.X (XX.X) | | | XX.X (XX.X) | | |
| Median | XX.X | | | XX.X | | |
| CV (%) | XX.X | | | XX.X | | |
| Q1, Q3 | XX.X, XX.X | | | XX.X, XX.X | | |
| Minimum, Maximum | XX.X, XX.X | | | XX.X, XX.X | | |
| sit 3/Week 4 | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV (%) | XX.X | - | - | XX.X | - | - |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| sit 5/Week 8 | | | | | | |
| N | XX | XX | XX | | | |
| <etc.></etc.> | | | | | | |

CFBL=Change from baseline; CV = Coefficient of Variation.

Note: Relative CFBL is defined as ratio of the post-baseline vs baseline value

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX / Reference: Data Listings XXXX

<Programming Note: Serum biochemistry tests include: cortisol, urea, glucose, creatinine, calcium, albumin, calcium (albumin corrected), sodium, potassium, chloride, calcium, phosphate, alkaline phosphatase (ALP), plasma parathyroid hormone (PTH). Hematology tests include: hemoglobin, hematocrit, red blood cell (RBC) count, mean corpuscular volume (MCV), white blood cell (WBC) count. Page break after each lab parameter.>

MC2 Therapeutics

Protocol Number: MC2-01-C3

Page X of Y

Table 14.3.2.2.X: Clinical Laboratory Results, Shifts from Baseline
[Biochemistry][Hematology]
Safety Population
[Lab Tests Name (Units)]

| | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) |
|---|---|---|
| Danking > Virit 2/(Varl. A (0/) | | |
| Baseline -> Visit 3/Week 4, n (%) | | |
| Low -> Normal | XX (XX.X) | XX(XX.X) |
| Normal -> Normal | XX (XX.X) | XX(XX.X) |
| High -> Normal | XX (XX.X) | XX(XX.X) |
| Normal -> Missing | XX (XX.X) | XX(XX.X) |
| Missing -> Low | XX (XX.X) | XX (XX.X) |
| <include all="" as="" possible="" rows="" shifts=""></include> | | |
| Baseline - > Most Extreme Post-Baseline Value up to Visit 3/Week 4, n (%) | | |
| Low -> Normal | XX (XX.X) | XX (XX.X) |
| Normal -> Normal | XX (XX.X) | XX (XX.X) |
| High -> Normal | XX (XX.X) | XX (XX.X) |
| Normal -> Missing | XX (XX.X) | XX (XX.X) |
| Missing -> Low | XX (XX.X) | XX (XX.X) |
| <include all="" as="" possible="" rows="" shifts=""></include> | , | ` , |

Note: Denominator is number of subjects with available baseline and post-baseline visit.

MC2 Therapeutics

Protocol Number: MC2-01-C3

Table 14.3.3: Summary of Vital Signs by Treatment and Visit
Safety Population
[Pulse Rate (bpm)][Systolic Blood Pressure (mmHg)][Diastolic Blood Pressure (mmHg)]

MC2-01 Cream (N=XX) Active Comparator (N=XX) **Observed Value Change from Baseline Observed Value Change from Baseline** Baseline XXXXΝ Mean (SD) XX (XX.X) XX (XX.X) Median XX (XX.X) XX (XX.X) Q1, Q3 XX, XX XX, XX Minimum, Maximum XX, XX XX, XX Visit 2/Week 2 N XXXX XXXXMean (SD) XX (XX.X) XX(XX.X)XX (XX.X) XX (XX.X) Median XX (XX.X) XX(XX.X)XX (XX.X) XX (XX.X) O1, O3 XX, XX XX, XX XX, XX XX, XX Minimum, Maximum XX, XX XX, XX XX, XX XX, XX Visit 3/Week 4 XXXXXXXXΝ Mean (SD) XX (XX.X) XX(XX.X)XX (XX.X) XX(XX.X)Median XX (XX.X) XX(XX.X)XX (XX.X) XX (XX.X) O1, O3 XX, XX XX, XX XX, XX XX, XX Minimum, Maximum XX, XXXX, XX XX, XX XX, XX <<Continue for all visits>>

Table 14.3.4: Summary of Investigator Assessed Local Skin Reactions (LSR)
Safety Population

| | MC2-01 Cream | Active Comparator |
|---|---|---|
| | (N=XX) | (N=XX) |
| Baseline | | |
| Perilesional Signs | | |
| Erythema, n(%) | | |
| N | XX | XX |
| 0 – Absent | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) |
| Severe Continue for Scaling, Edema, Atrophy, Vesicles, Erosion | | $M(M.\Lambda)$ |
| Continue for Searing, Edema, Attophry, Vesicles, Erosion | Olectation | |
| Lesional Signs | | |
| Vesicles, n(%) | | |
| N | XX | XX |
| 0 – None | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX (XX.X) | XX (XX.X) |
| 2 – Moderate | XX (XX.X) | XX (XX.X) |
| 3 – Severe | XX (XX.X) | XX (XX.X) |
| <continue erosion="" ulceration="">&gt;</continue> | ( ) | () |
| <continue all="" for="" visits="">&gt;</continue> | | |

Table 14.3.5: Summary of Subject Assessed Local Skin Reactions (LSR)
Safety Population

| | MC2-01 Cream<br>(N=XX) | Active Comparator (N=XX) |
|-----------------------|------------------------|--------------------------|
| | (2. 523) | (*) |
| Baseline | | |
| Burning or Pain, n(%) | | |
| N | XX | XX |
| 0 – Absent | XX (XX.X) | XX (XX.X) |
| 1 – Mild | XX(XX.X) | XX (XX.X) |
| 2 – Moderate | XX(XX.X) | XX (XX.X) |
| 3 – Severe | XX(XX.X) | XX (XX.X) |

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

Figure 14.4.1.1.X.Y: [CAL, BDP, MC1080, Betamethasone 17-propionate] Concentration (Median) by Time Point, Linear Scale [Week 4 Serial PK Sampling] [Week 8 Serial PK Sampling]

PK Population



[Time (hours)]

Note: Nominal sample collection times used in this figure. Concentrations below the limit of quantitation are reported as lower limit of quantification (LLOQ=XXXX).

Generated on XX/XX/XX XX:XX by XXXX / Uses: XXXX, XXXX, XXXX / Reference:

[Programming Note: include all time points pre-dose (0), 0.5, 1, 2, 3, 5, 7 Hour. The plot will include 2 lines (MC2-01 Cream and Active Comparator) at Week 4, 1 line (MC2-01 Cream) at Week 8.]

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

Figure 14.4.1.2.X.Y: [CAL, BDP, MC1080, Betamethasone 17-propionate] Concentration (Median) by Time Point, Semi-Log Scale [Week 4 Serial PK Sampling] [Week 8 Serial PK Sampling]

PK Population



[Time (hours)]

Note: Nominal sample collection times used in this figure. Concentrations below the limit of quantitation are reported as lower limit of quantification (LLOQ=XXXX).

Generated on XX/XX/XX XX:XX by XXXX / Uses: XXXX, XXXX, XXXX / Reference:

[Programming Note: include all time points pre-dose (0), 0.5, 1, 2, 3, 5, 7 Hour. The plot will include 2 lines (MC2-01 Cream and Active Comparator) at Week 4, 1 line (MC2-01 Cream) at Week 8.]

MC2 Therapeutics

Protocol Number: MC2-01-C3

Page X of Y

Figure 14.4.2.1.X.Y: Individual [CAL, BDP, MC1080, Betamethasone 17-propionate] Concentration (Median) by Time Point, Linear Scale

[Week 4 Serial PK Sampling] [Week 8 Serial PK Sampling]

PK Population

[MC2-01 Cream] [Active Comparator]

Subject: XXXX



[Time (hours)]

Note: Actual sample collection times used in this figure.

Generated on XX/XX/XX XX:XX by XXXX / Uses: XXXX, XXXX, XXXX / Reference:

[Programming Note: include all time points pre-dose (0), 0.5, 1, 2, 3, 5, 7 Hour.]

MC2 Therapeutics

Protocol Number: MC2-01-C3

Figure 14.4.2.2.X.Y: Individual [CAL, BDP, MC1080, Betamethasone 17-propionate] Concentration (Median) by Time Point, Semi-Log Scale

[Week 4 Serial PK Sampling] [Week 8 Serial PK Sampling]

PK Population

[MC2-01 Cream] [Active Comparator]

Subject: XXXX



[Time (hours)]

Note: Actual sample collection times used in this figure.

Generated on XX/XX/XX XX:XX by XXXX / Uses: XXXX, XXXX, XXXX / Reference:

[Programming Note: include all time points pre-dose (0), 0.5, 1, 2, 3, 5, 7 Hour.]

MC2 Therapeutics Protocol Number: MC2-01-C3

Data Listing 16.1.7: Subject Enrollment and Randomization All Randomized Subjects

| Subject<br>Number | Date of Informed<br>Consent | Require Washout<br>Period?/ Exclusion<br>Criteria | Washout Start<br>Date | Satisfy All<br>I/E Criteria? | Randomization<br>Date | Randomization<br>Number | Randomized<br>Treatment | Actual Treatment |
|---|---|---|---|---|---|---|---|---|
| XX-XXX | DDMMMYYYY | Yes / Exclusion X | DDMMYYYY | No: Inclusion XX | DDMMMYYYY | XXXX | MC2-01 Cream | MC2-01 Cream |
| XX-XXX | DDMMMYYYY | No | | Yes | DDMMMYYYY | XXXX | Active Comparator | Active Comparator |
| XX-XXX | DDMMMYYYY | No | | Yes | DDMMMYYYY | XXXX | MC2-01 Cream | Not Treated |

MC2 Therapeutics Protocol Number: MC2-01-C3

Data Listing 16.2.1.1: Screen Failures All Screen Failure Subjects

| Subject<br>Number | Date of Informed<br>Consent | Date of<br>Screening | Birth Month/Year | Age<br>(Years) | Sex | Primary Reason for<br>Screen Failure |
|---|---|---|---|---|---|---|
| XX-XXX | DDMMMYYYY | DDMMMYYYY | MMMYYYY | XX | X | I/E criteria not met: Inclusion 2 |
| XX-XXX | DDMMMYYYY | DDMMMYYYY | MMMYYYY | XX | X | Other: XXXXXXX |
| XX-XXX | DDMMMYYYY | DDMMMYYYY | MMMYYYY | XX | X | XXXXXXXXXX |
| XX-XXX | DDMMMYYYY | DDMMMYYYY | MMMYYYY | XX | X | XXXXXXXXXX |
| XX-XXX | DDMMMYYYY | DDMMMYYYY | MMMYYYY | XX | X | XXXXXXXXXX |

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

# Data Listing 16.2.1.2: Subject Disposition All Randomized Subjects [MC2-01 Cream][Active Comparator]

| | | | Dat | te (Day) of [1] | | | _ |
|---|---|---|---|---|---|---|---|
| Subject<br>Number | Screening | Randomization | First Dose | Last Dose | Last Visit | Last Contact | Completion<br>Status /<br>Discontinuation<br>Reason |
| XX-XXX<br>XX-XXX | ` ′ | , , | ` ′ | DDMMMYYYY(XX)<br>DDMMMYYYY(XX) | , , | ` ' | |
| 001-001 | 19JUN2017(-10) | 29JUN2017(1) | 29JUN2017(1) | | 06JUL2017(8) | | Completed |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

Data Listing 16.2.2: Protocol Deviation All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject<br>Number | Category | Major/Minor | Protocol Deviation |
|-------------------|----------|-------------|--------------------|
| XX-XXX | XXXX | Minor | xxxxxxxxxx |
| | XXXXX | Major | XXXX |

Generated on XX/XX/XX:XXXX by XXXX/ Uses: XXXX

<Programming Note: The format of protocol deviation listing depends on the actual protocol deviation report form layout. Additional columns may be added, such as "Reference" "Type". If site deviation or deviation for SF subjects are also available, include those at the very end of this listing.>

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

Data Listing 16.2.3: Population Datasets
All Randomized Subjects
[MC2-01 Cream][Active Comparator]

| Subject Number | In Safety Population? | In HDA Donulation? | In PK Population? | Reason for Exclusion from<br>Safety Population | Reason for Exclusion from HPA Population | Reason for Exclusion from PK Population |
|---|---|---|---|---|---|---|
| | in Salety Population: | In HFA Population: | In FK Population: | Safety Population | HEA POPULATION | rk ropulation |
| XX-XXX | Yes | Yes | No | NA | NA | XXX |
| XX-XXX | No | No | No | XXX | XXX | XXX |
| XX-XXX | XXX | XXX | XXX | NA | NA | NA |

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

# Data Listing 16.2.4.1: Demographics and Baseline Characteristics All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject<br>Number | Age (years) | Sex | Race | Ethnicity | Weight (kg) | Height (cm) | Fitzpatrick<br>Skin Type | HPA-axis<br>Suppression<br>Status[1] | PGA | Total BSA (%) | Duration of<br>Psoriasis<br>(years) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XX-XXX | XX | M | Asian | NH | XXX | XXX | X | Yes | X | XX.X | XX.X |
| XX-XXX | XX | F | White | Н | XXX | XXX | X | No | X | XX.X | XX.X |

Note: PGA = Physician's Global Assessment; BSA = Body Surface Area. NH=Not Hispanic or Latino; H=Hispanic or Latino [1] HPA-axis suppression status is only assessed among subjects assigned to MC2-01 cream.

### Data Listing 16.2.4.2: Prior and Concomitant Medication All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject<br>Number | Category | WHO Preferred Term<br>(Verbatim Term) /<br>ATC Classification | Topical treatment within 2 cm of treatment area?/ Indication Dose(Frequency)/Unit/Route | Administered for<br>AE #/ MH # | Start Date (Day)-Stop Date (Day) |
|---|---|---|---|---|---|
| XX-XXX | Prior | XXXXXX (xxxxx)/<br>XXXXXX | Yes/XXX<br>XX/XXX/XXXX | NA/1 | DDMMMYYYY (XX) –<br>DDMMMYYYY (XX) |
| XX-XXX | Concomitant | XXXXXX (xxxxx)/<br>XXXXXX | No/XXX<br>XX/XXX/XXXX | NA/NA | DDMMMYYYY (XX) –<br>Ongoing |

<sup>&</sup>lt;Programming Note: List medication in ascending start date for each subject.>

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

# Data Listing 16.2.4.3: Concurrent Procedures All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject Number | Preferred Term/<br>System Organ Class/<br>Procedure | Inside treatment area?/<br>Diagnosis/Body Location | Administered for<br>AE #/ MH # | Procedure Start Date (Day)-Stop Date (Day) |
|---|---|---|---|---|
| XX-XXX | XXXXXXX/<br>XXXXX/<br>XXXXXX | Yes/<br>XXXX/XXXXXXX | 1/NA | DDMMMYYYY (XX) – DDMMMYYYY (XX) |
| XX-XXX | XXXXXXX/<br>XXXXX/<br>XXXXXX | No/<br>XXXX/XXXXXXX | NA/NA | DDMMMYYYY (XX) – DDMMMYYYY (XX) |

<sup>&</sup>lt;Programming Note: List medication in ascending start date for each subject.>

MC2 Therapeutics

Protocol Number: MC2-01-C3

Page X of Y

#### Data Listing 16.2.4.4: Medical or Surgical History All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject Number | MH# | Diagnosis / Procedure | System Organ Class | Preferred Term | Ongoing? |
|---|---|---|---|---|---|
| XX-XXX | 1 | XXXX | XXXXX | XXXXXX | No |
| XX-XXX | 1 | XXXX | XXXXX | XXXXXX | Yes |

Data Listing 16.2.4.5: Psoriasis Treatment History
All Randomized Subjects
[MC2-01 Cream][Active Comparator]

| Subject<br>Number | Year of First Diagnosis of Psoriasis | Previous Treatment |
|---|---|---|
| XX-XXX | YYYY | TNF-a inhibitors |
| XX-XXX | YYYY | Topical: retinoids |

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

#### Data Listing 16.2.5.1: Study Drug Administration and Compliance All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject<br>Number | Visit | Visit Date (Day)[1] | Apply Study Drug<br>Once Daily Since Last Visit? | Number of<br>Missed Applications | Approved Stop Date (Day) [1] | Reason Missed |
|---|---|---|---|---|---|---|
| 3/3/ 3/3/3/ | 177 1 2/117 1 2 | | ** | 3/3/ | 27.4 | 27.4 |
| XX-XXX | Visit 2/Week 2 | DDMMMYYYY(XX) | Y | XX | NA | NA |
| | Visit 3/Week 4 | DDMMMYYYY(XX) | Y | XX | NA | NA |
| | Visit 4/Week 6 | DDMMMYYYY(XX) | Y | XX | NA | NA |
| | Visit 5/Week 8 | DDMMMYYYY(XX) | N | XX | DDMMMYYYY(XX) | XXXXXXXXXX |
| XX-XXX | Visit 2/Week 2 | DDMMMYYYY(XX) | Y | XX | NA | NA |
| | Visit 3/Week 4 | DDMMMYYYY(XX) | Y | XX | NA | NA |
| | Visit 4/Week 6 | DDMMMYYYY(XX) | N | XX | NA | NA |
| | Visit 5/Week 8 | DDMMMYYYY(XX) | N | XX | DDMMMYYYY(XX) | XXXXXXX |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

Data Listing 16.2.5.2: Study Drug Accountability
All Randomized Subjects
[MC2-01 Cream][Active Comparator]

| Subject<br>Number | Visit | Kit Number | Date (Day)<br>Dispensed [1] | Tube Number | Tube Retuned? | Date (Day) Returned [1] | Tube Sealed? | Return Weight (g) |
|---|---|---|---|---|---|---|---|---|
| Tumber | VISIT | Kit Ivallibei | Dispenseu [1] | Tube Number | Tube Retuneu. | Date (Day) Returned [1] | Tube Scarcu. | Return Weight (g) |
| XX-XXX | Visit 1/Day 1 | XXXXXXX | DDMMMYYYY(XX) | 1 | Yes | DDMMMYYYY(XX) | XX | XX.X |
| | | | | 2 | No | DDMMMYYYY(XX) | - | - |
| | Visit 2/Week 2 | XXXXXXX | DDMMMYYYY(XX) | 1 | Yes | DDMMMYYYY(XX) | XX | XX.X |
| | | | | 2 | Redispensed | - | - | - |
| | Visit 3/Week 4 | XXXXXXX | DDMMMYYYY(XX) | 1 | XXXX | DDMMMYYYY(XX) | XX | XX.X |
| | | | | 2 | XXXX | DDMMMYYYY(XX) | XX | XX.X |
| XX-XXX | Visit 1/Day 1 | XXXXXXX | DDMMMYYYY(XX) | 1 | Redispensed | DDMMMYYYY(XX) | XX | XX.X |
| | | | | 2 | No | DDMMMYYYY(XX) | XX | XX.X |
| | Visit 2/Week 2 | XXXXXXX | DDMMMYYYY(XX) | 1 | Yes | DDMMMYYYY(XX) | XX | XX.X |
| | | | | 2 | Redispensed | DDMMMYYYY(XX) | XX | XX.X |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

### Data Listing 16.2.5.3.1: Overall Study Drug Exposure and Compliance, Day 1 to Week 4 Period All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject<br>Number | Total Number of Days of Exposure[1] | Total Number of<br>Expected Doses[2] | Total Number of<br>Missed Doses | Total Number of<br>Applied Doses[3] | Total Amount of Drug<br>Used (g)[4] | Amount of Drug Used per<br>week (g/per week)[5] |
|---|---|---|---|---|---|---|
| XX-XXX | XX | XX | XX | XX | XX.X | XX.X |
| XX-XXX | XX | XX | XX | XX | XX.X | XX.X |

<sup>[1]</sup> Total number of days of exposure to the study drug is defined as the date of last application of study drug minus date of first application plus one. Last application is applied in-clinic at Week 4 visit.

<sup>[2]</sup> Total number of expected doses is defined as total number of days of exposure minus any days of investigator approved stop (if applicable)

<sup>[3]</sup> Total number of doses applied, defined as the total number of doses required minus total number of doses missed.

<sup>[4]</sup> Total amount of drug used (g), defined as the summation of amount of drug used per kit for all dispensed kits.

<sup>[5]</sup> Amount of drug used per week (g/per week), defined as the total amount of drug used divided by total number of days of exposure to the study drug multiplied by 7.

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

Data Listing 16.2.5.3.2: Overall Study Drug Exposure and Compliance, Day 1 to Week 8 Period All Randomized Subjects

[MC2-01 Cream]

| Subject<br>Number | Total Number of Days of Exposure[1] | Total Number of<br>Expected Doses[2] | Total Number of<br>Missed Doses | Total Number of<br>Applied Doses[3] | Total Amount of Drug<br>Used (g)[4] | Amount of Drug Used per<br>week (g/per week)[5] |
|---|---|---|---|---|---|---|
| XX-XXX | XX | XX | XX | XX | XX.X | XX.X |
| XX-XXX | XX | XX | XX | XX | XX.X | XX.X |

<sup>[1]</sup> Total number of days of exposure to the study drug is defined as the date of last application of study drug minus date of first application plus one. Last application is applied in-clinic at Week 8 visit.

<sup>[2]</sup> Total number of expected doses is defined as total number of days of exposure minus any days of investigator approved stop (if applicable)

<sup>[3]</sup> Total number of doses applied, defined as the total number of doses required minus total number of doses missed.

<sup>[4]</sup> Total amount of drug used (g), defined as the summation of amount of drug used per kit for all dispensed kits.

<sup>[5]</sup> Amount of drug used per week (g/per week), defined as the total amount of drug used divided by total number of days of exposure to the study drug multiplied by 7.

MC2 Therapeutics

Protocol Number: MC2-01-C3

Data Listing 16.2.5.4.1: Subject Treatment Diary Card All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject | | | |
|---|---|---|---|
| Number | Date (Day)[1] | Study Drug Applied? | Reason if Medication not Applied |
| XX-XXX | DDMMMYYYY (1) | Y | - |
| | DDMMMYYYY (XX) | Y | - |
| | DDMMMYYYY (XX) | N | XXXXXXX |

[1] Study day is calculated relative to date of first application of study drug (Day 1).

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

#### Data Listing 16.2.5.4.2: Subject Food Diary All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject | | | | Number of Servings of | • |
|---|---|---|---|---|---|
| Number | Visit | Time Point | Date (Day)[1] | Calcium-rich Foods | Reason Not Done |
| XX-XXX | Visit 1/Day 1 | Day -3 | DDMMMYYYY (-3) | X | NA |
| | Visit 1/Buy 1 | Day -2 | DDMMMYYYY (-2) | X | NA |
| | | Day -1 | DDMMMYYYY (-1) | X | XXXXXXX |
| | | Collection Day | DDMMMYYYY (1) | | |

[1] Study day is calculated relative to date of first application of study drug (Day 1).

Listing 16.2.6.1: Plasma Concentration Sample Date and Time and Plasma Concentrations
PK Population
[MC2-01 Cream] [Active Comparator]

| Subject | Visit | Dosing Date and Time | PK Time Point | Sample Collection Date and<br>Time (Day) | Elapsed<br>Time<br>(hours) | CAL<br>(unit) | BDP<br>(unit) | MC1080<br>(unit) | Betamethasone<br>17-propionate<br>(unit) |
|---|---|---|---|---|---|---|---|---|---|
| XX-<br>XXX | Baseline | | | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Visit 2/<br>Week 2 | DDMMYYYYTXX:XX | Pre-dose | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Visit 3/<br>Week 4 | DDMMYYYYTXX:XX | Pre-dose | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | 0.5 hour post-<br>dose | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | 1 hour post-dose | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | 2 hours post-dose | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | 3 hours post-dose | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | 5 hours post-dose | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | 7 hours post-dose <etc.></etc.> | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Visit 5/<br>Week 8 | DDMMYYYYTXX:XX | Pre-dose | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | 0.5 hour post-<br>dose<br><etc.></etc.> | DDMMYYYYTXX:XX (XX) | XX.X | XX.X | XX.X | XX.X | XX.X |

MC2 Therapeutics

Protocol Number: MC2-01-C3

Listing 16.2.6.2.X: [CAL, BDP, MC1080, Betamethasone 17-propionate] Derived Pharmacokinetics Parameters PK Population
[MC2-01 Cream] [Active Comparator]

| XXX-XXX Week 4 XXXX XXXX XXXXX XXXXX XXXXX XX | Subject | Visit | C <sub>max</sub> (ng/mL) | T <sub>max</sub> (h) | AUC <sub>0-7</sub> (ng*h/mL) | AUC <sub>0-t</sub> (ng*h/mL) | AUC₀-∞ (ng*h/mL) | $T_{1/2}$ (h) |
|---|---|---|---|---|---|---|---|---|
| | XXX-XXX | Week 4 | XXXX | XXXX | XX.XX | XXXXX | XXXXX | XXXX |
| Week 8 XXXX XXXX XXXXX XXXXX XXXXX XXXXX XX | | Week 8 | XXXX | XXXX | XX.XX | XXXXX | XXXXX | XXXX |

Generated on XX/XX/XX:XXXX by XXXX / Uses: XX

[Programming Note: Week 8 only applies to MC2-01 Cream subjects]

MC2 Therapeutics

Protocol Number: MC2-01-C3

Data Listing 16.2.6.3: Physician's Global Assessment of Disease Severity (PGA) – Scalp, Trunk and/or Limbs All Randomized Subjects
[MC2-01 Cream][Active Comparator]

| Subject Number | Visit | Visit Date (Day) [1] | PGA | Change from Baseline | Treatment<br>Success?[2] |
|---|---|---|---|---|---|
| XX-XXX | Screening | DDMMMYYYY(XX) | 3 – Moderate | | |
| | Visit 1/Day 1 | DDMMMYYYY(XX) | 3 – Moderate | | |
| | Visit 2/Week 2 | DDMMMYYYY(XX) | 2 - Mild | -1 | N |
| | Visit 3/Week 4 | DDMMMYYYY(XX) | 2 – Mild | -1 | N |
| | Visit 4/Week 6 | DDMMMYYYY(XX) | 1 – Almost clear | -2 | Y |
| | Visit 5/Week 8 | DDMMMYYYY(XX) | 1 – Almost clear | -2 | Y |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

<sup>[2]</sup> PGA success is defined as a minimum 2-point decrease from Baseline in the PGA.

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

Data Listing 16.2.6.4: Investigator's Assessment of the Body Surface Area (BSA) Involvement of Psoriasis
All Randomized Subjects
[MC2-01 Cream][Active Comparator]

| Subject<br>Number | Visit | Visit Date (Day) [1] | Scalp BSA (%) | Neck, Trunk and/or Limbs BSA (%) | Total BSA (%) |
|---|---|---|---|---|---|
| XX-XXX | Screening | DDMMMYYYY(XX) | XX.X | XX.X | XX.X |
| | Visit 1/Day 1 | DDMMMYYYY(XX) | XX.X | XX.X | XX.X |
| | Visit 3/Week 4 | DDMMMYYYY(XX) | XX.X | XX.X | XX.X |
| | Visit 5/Week 8 | DDMMMYYYY(XX) | XX.X | XX.X | XX.X |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

Data Listing 16.2.6.5: Investigator and Subject Assessed Local Skin Reaction (LSR)
All Randomized Subjects
[MC2-01 Cream][Active Comparator]

| | | | Investigator Assessed | | | | | | Subject<br>Assessed | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Visit | sit Visit Date (Day) [1] | Perilesional Signs | | | Lesional Signs | | | | Burning or | |
| | | | Erythema | Scaling | Edema | Atrophy | Vesicles | Erosion/<br>Ulceration | Vesicles | Erosion/<br>Ulceration | Pain Pain |
| XX-XXX | Visit 1/Day 1 | DDMMMYYYY(XX) | 1=Mild | 1=Mild | 1=Mild | 3=Severe | X | X | X | X | X |
| | Visit 2/Week 2 | DDMMMYYYY(XX) | X | X | X | X | X | X | X | X | X |
| | Visit 3/Week 4 | DDMMMYYYY(XX) | X | X | X | X | X | X | X | X | X |
| | Visit 4/Week 6 | DDMMMYYYY(XX) | X | X | X | X | X | X | X | X | X |
| | Visit 5/Week 8 | DDMMMYYYY(XX) | X | X | X | X | X | X | X | X | X |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

### Data Listing 16.2.6.6: Psoriasis Treatment Convenience Scale All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject Number | Visit | Visit Date (Day) [1] | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Total Score of Q1-Q5 |
|---|---|---|---|---|---|---|---|---|---|
| XX-XXX | Visit 3/Week 4 | DDMMMYYYY(XX) | XX | XX | XX | XX | XX | XX | XX |
| XX-XXX | Unscheduled | DDMMMYYYY(XX) | XX | XX | XX | XX | XX | XX | XX |

Q1 = How easy was the treatment to apply to the skin?; Q2 = How greasy was the treatment when applying it to the skin?; Q3 = How moisturized did your skin feel after applying the treatment?; Q4 = How greasy did your skin feel after applying the treatment?; Q5 = How much did treating your skin disrupt your daily routine?; Q6 = Overall, how satisfied were you with the medical treatment?

[1] Study day is calculated relative to date of first application of study drug (Day 1).
MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

#### Data Listing 16.2.6.7: ACTH Challenge All Randomized Subjects [MC2-01 Cream][Active Comparator]

| | | | | Pre-Stin | nulation | 30 Min Po | ost-Stimulation | <b>HPA-Axis</b> |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Visit | Date (Day) [1] | Cosyntropin<br>Injection Time | <b>Collection Time</b> | Cortisol Level<br>(µg/dL) | Collection Time | Cortisol Level<br>(µg/dL) | Suppression |
| XX-XXX | Visit 1/Day 1 | DDMMMYYYY (XX) | HH:MM | HH:MM | XX.X | HH:MM | XX.X | No |
| | Visit 3/Week 4 | DDMMMYYYY (XX) | HH:MM | HH:MM | XX.X | HH:MM | XX.X | No |
| | Visit 4/Week 8 | DDMMMYYYY (XX) | HH:MM | HH:MM | XX.X | HH:MM | XX.X | Yes |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

Page X of Y

MC2 Therapeutics

Protocol Number: MC2-01-C3

Data Listing 16.2.7.1: Adverse Events All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject AE<br>Number # | MedDRA SOC Term/<br>MedDRA Preferred<br>Term /<br>(Verbatim Term) | TEAE? [1] / Period<br>Onset Date (Day) –<br>End Date (Day) [2] | Related to<br>Cosyntropin?/<br>Related to Study<br>Procedure? | Outcome/<br>Withdraw due to<br>AE? | SAE: Criteria?/<br>Severity | Location to Treatment<br>Area/<br>Relationship to Study<br>Medication | Action Taken /<br>Other Action<br>Taken |
|---|---|---|---|---|---|---|---|
| XX-XXX 1 | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | Yes / 1<br>DDMMMYYYY(XX) –<br>DDMMMYYYY(XX) | No/No | XXXXXXXX/<br>Yes | Yes:<br>Hospitalization /<br>Mild | Inside treatment area/<br>Definitely Related | XXXXXXXX /<br>XXXXXXXX |
| 2 | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | No / NA<br>DDMMMYYYY(XX) –<br>Ongoing | No/Yes | XXXXXXX/<br>No | No/<br>XXXXXXXX | Outside treatment area/<br>XXXXXXXX | XXXXXXXX /<br>XXXXXXXX |
| XX-XXX 1 | XXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | Yes / 2<br>DDMMMYYYY(XX) –<br>DDMMMYYYY(XX) | No/No | XXXXXXXX/<br>XX | No/<br>XXXXXXXX | Non-cutaneous/<br>XXXXXXXX | XXXXXXXX /<br>XXXXXXXX |

Period 1=Week 1-4; Period 2=Post Week4.

Generated on XX/XX/XX:XXXX by LSTAE / Uses: AE

<sup>[1]</sup> A treatment-emergent AE (TEAE) is defined as an AE with a start date on or after the first application to trial medication.

<sup>[2]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

#### Data Listing 16.2.7.2: Serious Adverse Events All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject AE<br>Number # | MedDRA SOC Term/<br>MedDRA Preferred<br>Term /<br>(Verbatim Term) | TEAE? [1] / Period<br>Onset Date (Day) –<br>End Date (Day) [2] | Related to<br>Cosyntropin?/<br>Related to Study<br>Procedure? | Outcome/<br>Withdraw due to<br>AE? | SAE Criteria/<br>Severity | Location to Treatment<br>Area/<br>Relationship to Study<br>Medication | Action Taken /<br>Other Action<br>Taken |
|---|---|---|---|---|---|---|---|
| XX-XXX 1 | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | Yes / 1<br>DDMMMYYYY(XX) –<br>DDMMMYYYY(XX) | No/No | XXXXXXXX/<br>Yes | Hospitalization /<br>Mild | Inside treatment area/<br>Definitely Related | XXXXXXXX /<br>XXXXXXXX |
| XX-XXX 2 | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | No / NA<br>DDMMMYYYY(XX) –<br>DDMMMYYYY(XX) | No/No | XXXXXXXX/<br>No | XXX/<br>XXXXXXXX | Non-cutaneous/<br>XXXXXXXX | XXXXXXXX /<br>XXXXXXXX |

Period 1=Week 1-4; Period 2=Post Week4.

Generated on XX/XX/XX:XXXX by LSTAE / Uses: AE

<sup>[1]</sup> A treatment-emergent AE (TEAE) is defined as an AE with a start date on or after the first application to trial medication.

<sup>[2]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

# Data Listing 16.2.7.3: Adverse Events Leading to Study Drug Discontinuation All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject<br>Number | AE<br># | MedDRA SOC Term/<br>MedDRA Preferred<br>Term/<br>(Verbatim Term) | TEAE? [1] / Period<br>Onset Date (Day) –<br>End Date (Day) [2] | Related to<br>Cosyntropin?/<br>Related to Study<br>Procedure? | Outcome/<br>Withdraw due to<br>AE? | SAE: Criteria?/<br>Severity | Location to Treatment<br>Area/<br>Relationship to Study<br>Medication | Other Action<br>Taken |
|---|---|---|---|---|---|---|---|---|
| XX-XXX | 1 | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | Yes / 1<br>DDMMMYYYY(XX) –<br>DDMMMYYYY(XX) | No/No | XXXXXXXX/<br>Yes | Yes:<br>Hospitalization /<br>Mild | Inside treatment area/<br>Definitely Related | XXXXXXX |
| | 2 | XXXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | No / NA<br>DDMMMYYYY(XX) –<br>Ongoing | No/Yes | XXXXXXX/<br>No | No/<br>XXXXXXXX | Outside treatment area/<br>XXXXXXXX | XXXXXXX |
| XX-XXX | 1 | XXXXXXX /<br>XXXXXXXX /<br>(XXXXXXXX) | Yes / 2<br>DDMMMYYYY(XX) –<br>DDMMMYYYY(XX) | No/No | XXXXXXXX/<br>XX | No/<br>XXXXXXXX | Non-cutaneous/<br>XXXXXXXX | XXXXXXX |

Period 1=Week 1-4; Period 2=Post Week4.

Generated on XX/XX/XX:XXXX by LSTAE / Uses: AE

<sup>[1]</sup> A treatment-emergent AE (TEAE) is defined as an AE with a start date on or after the first application to trial medication.

<sup>[2]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

MC2 Therapeutics

Protocol Number: MC2-01-C3

Page X of Y

# Data Listing 16.2.8.1: Urine Pregnancy Test All Randomized Female Subjects with Childbearing Potential [MC2-01 Cream][Active Comparator]

| Number | Birth Control Methods | Visit | Date of Test (Day)[1] | Result |
|---|---|---|---|---|
| XX-XXX | Abstinence | Screening | DDMMMYYYY(XX) | Negative |
| | | Visit 1/Day 0 | DDMMMYYYY(XX) | Negative |
| | | Visit 3/Week 4 | DDMMMYYYY(XX) | Negative |
| | | Visit 5/Week 8 | DDMMMYYYY(XX) | Negative |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

Generated on XX/XX/XX:XXXX by XXXX / Uses: XX

MC2 Therapeutics Page X of Y

Protocol Number: MC2-01-C3

# Data Listing 16.2.8.2.X: Clinical Laboratory Test [Biochemistry][Hematology] All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject<br>Number | Visit | Date (Day) and Time of Sample[1] | Parameter (Unit) | Reference Range | Results | Abnormality | CFBL |
|---|---|---|---|---|---|---|---|
| XX-XXX | Visit 1/Day 1 | DDMMMYYYY (XX)THH:MM | XXXX | XXXX,XXXX | XX.XX | | |
| | | | XXXX | XXXX,XXXX | XX.XX | High | |
| | | | XXXX | XXXX,XXXX | XX.XX | | XXX.X |
| | Visit 3/Week 4 | DDMMMYYYY (XX) | XXXX | XXXX,XXXX | XX.XX | Low | XXX.X |
| | Visit 4/Week 8 | DDMMMYYYY (XX) | XXXX | XXXX,XXXX | XX.XX | | XXX.X |

CFBL = Change from Baseline

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

Page X of Y

MC2 Therapeutics

Protocol Number: MC2-01-C3

Data Listing 16.2.8.2.3: Clinical Laboratory Test 24 Hour Urinalysis All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject<br>Number | Visit | Collection Date and Time<br>Start – Stop | Total Volume<br>Collected (mL) | Parameter<br>(Unit) | Reference Range | Results | Abnormality | CFBL |
|---|---|---|---|---|---|---|---|---|
| | | DDMMYYYY(DD)THH:MM- | | | | | | |
| XX-XXX | Visit 1/Day 1 | DDMMYYYY(DD)THH:MM | XXXX | XXXX | XXXX,XXXX | XX.XX | | |
| | | | | XXXX | XXXX,XXXX | XX.XX | High | |
| | | | | XXXX | XXXX,XXXX | XX.XX | | XXX.X |
| | Visit 3/Week 4 | | | XXXX | XXXX,XXXX | XX.XX | Low | XXX.X |
| | Visit 4/Week 8 | | | XXXX | XXXX,XXXX | XX.XX | | XXX.X |

CFBL = Change from Baseline

[1] Study day is calculated relative to date of first application of study drug (Day 1).

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX

[Programming Note: Week 4 and Week 8 only applies to MC2-01 Cream subjects]

MC2 Therapeutics

Protocol Number: MC2-01-C3

Page X of Y

#### Data Listing 16.2.8.3: Laboratory Values Outside of Normal Range All Randomized Subjects [MC2-01 Cream][Active Comparator]

| Subject Number | Visit | Date (Day) of Sample[1] | Category | Parameter (Unit) | Reference Range | Results | Abnormality | CFBL |
|---|---|---|---|---|---|---|---|---|
| XX-XXX | Visit 1/Day 1 | DDMMMYYYY (XX) | Biochemistry | XXXX | XXXX,XXXX | XX.XX | High | |
| | | | Hematology | XXXX | XXXX,XXXX | XX.XX | High | |
| | | | Urinalysis | XXXX | XXXX,XXXX | XX.XX | | XXX.X |
| | Visit 3/Week 4 | DDMMMYYYY (XX) | | XXXX | XXXX,XXXX | XX.XX | Low | XXX.X |
| | Visit 4/Week 8 | DDMMMYYYY (XX) | | XXXX | XXXX,XXXX | XX.XX | | XXX.X |

CFBL = Change from Baseline

Generated on XX/XX/XX:XXXX by XXXXX / Uses: XX

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

Page X of Y

MC2 Therapeutics

Protocol Number: MC2-01-C3

Data Listing 16.2.8.4: Vital Signs All Randomized Subjects [MC2-01 Cream][Active Comparator]

| 6.11 | | | SBP (n | nmHg) | DBP (n | nmHg) | Pulse Ra | ate (bpm) |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Visit | Visit Date (Day) [1] | Observed | CFBL | Observed | CFBL | Observed | CFBL |
| XX-XXX | Screening | DDMMYYYY (XX) | XX.X | | XX.X | | XX.X | |
| | Visit 1/Day 1 | DDMMYYYY (XX) | XX.X | | XX.X | | XX.X | |
| | Visit 2/Week 2 | DDMMYYYY (XX) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Visit 3/Week 4 | DDMMYYYY (XX) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Visit 4/Week 6 | DDMMYYYY (XX) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Visit 5/Week 8 | DDMMYYYY (XX) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Note: SBP=Systolic blood pressure; DBP=Diastolic blood pressure; CFBL= change from baseline

[1] Study day is calculated relative to date of first application of study drug (Day 1).

Generated on XX/XX/XX:XXXX by XXXX / Uses: XXXX

MC2 Therapeutics
Page X of Y
Protocol Number: MC2-01-C3

Data Listing 16.2.8.5: Physical Examination Randomized Subjects with Abnormal Results [MC2-01 Cream][Active Comparator]

| Subject<br>Number | Visit | Visit Date (Day) [1] | Findings |
|---|---|---|---|
| XX-XXX | Screening | DDMMMYYYY (XX) | Abnormal Not Clinically Significant |
| XX-XXX | XXXX | DDMMMYYYY (XX) | Abnormal Clinically Significant |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

MC2 Therapeutics Protocol Number: MC2-01-C3 Page X of Y

Data Listing 16.2.8.6: 12-Lead ECG Results
All Randomized Subjects
[MC2-01 Cream][Active Comparator]

| Subject<br>Number | Visit | Visit Date (Day) [1] | ECG Test (Units) | Result |
|---|---|---|---|---|
| XX-XXX | Visit 1/Day 1 | DDMMMYYYY (XX) | Interpretation | Abnormal Not Clinically Significant |
| | | DDMMMYYYY (XX) | ECG Finding 1 | XXXXX |
| | | DDMMMYYYY (XX) | ECG Finding 2 | XXXX |
| | | | Summary (Mean) Heart Rate (b | peats/min) |
| | | | Summary (Mean) RR Duration | (msec) |
| | | | Etc. | |
| | Visit 3/Week 4 | DDMMMYYYY (XX) | XXXXX | XXXXX |
| | Visit 5/Week 8 | DDMMMYYYY (XX) | XXXXX | XXXXX |

<sup>[1]</sup> Study day is calculated relative to date of first application of study drug (Day 1).

Generated on XX/XX/XX:XXXX by LSTEG/ Uses: XXXX

MC2 Therapeutics Protocol No. MC2-01-C3 Novella No. NYA14539

 September 20, 2018

MC2 Therapeutics Protocol Number: MC2-01-C3

Page X of Y

Data Listing 16.2.9: General Comments [MC2-01 Cream][Active Comparator]

| Subject | | |
|---------|--------------------------|-----------------------------------------|
| Number | <b>Comment Reference</b> | Comment |
| XX-XXX | Visit 3/Week 4 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XX-XXX | Visit 5/Week 8 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |



**Certificate Of Completion** 

Envelope Id: C72CEACD45E649FEBAEF9862708CB5E6

Subject: Please DocuSign: MC2-01-C3 SAP 21sep2018 Amendment 1 clean.pdf

Source Envelope:

Document Pages: 84 Signatures: 2 **Envelope Originator:** 

Initials: 0 jin Wei Certificate Pages: 5 1700 Perimeter Park Drive

AutoNav: Enabled

Envelopeld Stamping: Disabled Morrisville, NC 27560 Time Zone: (UTC-05:00) Eastern Time (US & Canada) Jin.Wei2@novellaclinical.com

IP Address: 192.69.83.249

Signed: 9/21/2018 12:15:46 PM

Status: Completed

**Record Tracking** 

Status: Original Holder: iin Wei Location: DocuSign

9/21/2018 11:36:32 AM Jin.Wei2@novellaclinical.com

**Signature Timestamp** Signer Events Carol Udell Sent: 9/21/2018 11:40:43 AM Carol Udell Carol.Udell@novellaclinical.com Viewed: 9/21/2018 12:13:46 PM

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

CE741CD0-FE97-41EC-A29C-B39E84B183BB

Using IP Address: 192.69.82.248

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 6/29/2017 9:05:59 AM

ID: 23a67abb-661c-48d7-a3b0-5cd8fbe94ff5

Johan Selmer

jse@mc2therapeutics.com

Security Level: Email, Account Authentication

(Required)

Johan Selmer

Sent: 9/21/2018 11:40:43 AM Viewed: 9/21/2018 11:42:51 AM

Signed: 9/21/2018 11:43:37 AM

Signature Adoption: Pre-selected Style

Signature ID:

0CB84AC3-A754-477D-9A78-70027DF16AE6

Using IP Address: 77.72.48.114

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): Jeg godkender dette dokument

**Electronic Record and Signature Disclosure:** 

Accepted: 5/16/2018 6:58:25 AM

ID: 7622460b-6a54-44da-884b-23e798fe761d

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |

**Carbon Copy Events** 

Birgitte Vestbjerg

bve@mc2therapeutics.com

Security Level: Email, Account Authentication

(Required)

**Electronic Record and Signature Disclosure:** 

Accepted: 8/21/2017 9:01:36 AM

ID: 2f1c7a3f-d74e-4f4c-b2f9-9471674f2918

Status **Timestamp** 

**COPIED** 

Sent: 9/21/2018 11:40:44 AM

| Notary Events | Signature | Timestamp |
|-------------------------|------------------|-----------------------|
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 9/21/2018 11:40:44 AM |
| Certified Delivered | Security Checked | 9/21/2018 12:13:47 PM |
| Signing Complete | Security Checked | 9/21/2018 12:15:46 PM |
| Completed | Security Checked | 9/21/2018 12:15:46 PM |
| Payment Events | Status | Timestamps |

**Electronic Record and Signature Disclosure** 

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Novella Clinical DocuSign Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

# Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# **How to contact Novella Clinical DocuSign Part 11:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: ngliatis@novellaclinical.com

#### To advise Novella Clinical DocuSign Part 11 of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at ngliatis@novellaclinical.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

## To request paper copies from Novella Clinical DocuSign Part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to ngliatis@novellaclinical.com and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with Novella Clinical DocuSign Part 11

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to ngliatis@novellaclinical.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| 1 | |
|----------------------------|----------------------------------------------|
| Operating Systems: | Windows2000? or WindowsXP? |
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | -Anow per session cookies |
| | •Users accessing the internet behind a Proxy |
| | Server must enable HTTP 1.1 settings via |
| | proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

#### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Novella Clinical DocuSign Part 11 as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Novella Clinical DocuSign Part 11 during the course of my relationship with you.